### elMPACT Trial:

# Modernized Collaborative Care to Reduce the Excess CVD Risk of Older Depressed Patients

(ClinicalTrials.gov ID: NCT02458690)

# Trial Protocol 7/13/2018

# Jesse C. Stewart, Ph.D.

Principal Investigator
Department of Psychology
Indiana University-Purdue University Indianapolis
402 N. Blackford Street, LD 100E
Indianapolis, IN 46202

# Christopher M. Callahan, M.D.

Co-Investigator
Department of Medicine
Indiana University School of Medicine
HITS Suite 2000
Indianapolis, IN 46202

# John I. Nurnberger, Jr., M.D., Ph.D.

Co-Investigator
Department of Psychiatry
Indiana University School of Medicine
791 Union Drive
Indianapolis, IN 46202

# Samir K. Gupta, M.D., M.S.

Co-Investigator
Department of Medicine
Indiana University School of Medicine
Emerson Hall, Room 421
545 N. Barnhill Dr.
Indianapolis, IN 46202-5124

### Richard J. Kovacs, M.D.

Co-Investigator
Department of Medicine
Indiana University School of Medicine
Krannert Institute of Cardiology, Room E300
1801 N. Senate Blvd., Suite E4000
Indianapolis, IN 46202

# Robert V. Considine, Ph.D.

Co-Investigator
Department of Medicine
Indiana University School of Medicine
Gatch Clinical Building, Room 455
1120 W. Michigan Street
Indianapolis, IN 46202

# Sujuan Gao, Ph.D.

Co-Investigator
Department of Biostatistics
Indiana University School of Medicine
410 West 10th Street, Suite 3000
Indianapolis, IN 46202

# Bruce L. Rollman, M.D., M.P.H.

Consultant

Professor of Medicine, Psychiatry,
Clinical and Translational Sciences, and Biomedical Informatics
University of Pittsburgh School of Medicine
230 McKee Place, Suite 600
Pittsburgh, PA 15213

### **Table of Contents:**

# **Study Schema**

- 1.0 Background
- 2.0 Rationale and Specific Aims
- 3.0 Inclusion/Exclusion Criteria
- 4.0 Enrollment/Randomization
- 5.0 Study Procedures
- 6.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 7.0 Study Withdrawal/Discontinuation
- 8.0 Statistical Considerations
- 9.0 Privacy/Confidentiality Issues
- 10.0 Follow-Up and Record Retention

# 1.0 Background

# **Significance**

CVD and depression are top public health concerns; they are highly prevalent, deadly, and costly. CVD is highly prevalent and disproportionately affects older adults.<sup>1</sup> A total of 15.4 and 6.8 million Americans suffer from coronary artery disease (CAD) and cerebrovascular disease (CBV).<sup>1</sup> CVD is also deadly. CAD and CBV are the first and fourth leading causes of death in the U.S.<sup>2</sup> Finally, the economic burden of CVD is substantial. For 2009, total cost in the U.S. was estimated to be \$312.6 billion, which is greater than all cancers.<sup>1</sup> Furthermore, due to the rapidly growing elderly population, the prevalence of CAD and CBV are projected to increase by 18-22% by 2030, and the total cost is expected more than double.<sup>1</sup>

Depression is also a top concern. In the U.S., major depressive disorder (MDD) has a lifetime prevalence of 16.2%,<sup>3</sup> and the point prevalence of depressive disorders in primary care is 16-19%.<sup>4,5</sup> Depression is the leading cause of disability,<sup>6</sup> and the annual total cost of depression is over \$83.1 billion.<sup>7</sup> By 2020, CVD and depression are projected to be the #1 and #2 causes of disease burden worldwide.<sup>6</sup>

# Depression is an independent risk and prognostic factor for CVD.

Thirty years of evidence indicates that depression is an independent risk and prognostic factor for CAD and CBV.<sup>8,9</sup> Meta-analyses have shown that adults with a depressive disorder or symptoms have a 64% greater risk of CAD onset<sup>10,11</sup> and that depressed CAD patients have a 59% greater likelihood of a future CVD event than their nondepressed counterparts.<sup>9</sup> The depression-CVD relationship is comparable in strength to conventional CVD risk factors<sup>12</sup> and has been detected in men and women and in various age and racial/ethnic groups.<sup>8,13-15</sup> Although other emotional factors have been linked to CVD,<sup>16</sup> the depression association is the most consistently observed<sup>16</sup> and seems to be independent of anxiety and hostility/anger.<sup>17</sup> CVD risk increases with depression severity,<sup>10</sup> indicating a dose-response relationship. Finally, depression has been linked to several atherogenic factors, which supports the biological plausibility of these prospective associations.

Because depression satisfies 8 of Hill's 9 criteria for causation,<sup>18</sup> it is reasonable to conclude that depression is an independent, and potentially causal, risk factor for CVD. Experimental animal research also supports a causal relationship between depression and atherogenesis.<sup>19</sup> The lack of experimental evidence in humans, however, prevents one from drawing a causal inference, as the possibility that a third factor (e.g., genetic variants related to inflammation) explains the depression-CVD association has not been ruled out.<sup>20</sup>

The Problem: Attempts to improve CVD outcomes of depressed patients have been unsuccessful. Despite this strong evidence base, the few trials that have evaluated whether depression interventions reduce the likelihood of CVD events generally have not observed the anticipated benefits. A key study was the Enhancing Recovery in Coronary Heart Disease (ENRICHD) Patients trial, in which 2,481 post-MI patients with depression and/or low social support were randomized to cognitive-behavioral therapy (CBT) or usual care. After 29 months, no difference in nonfatal MI or death was found. 21 In the Sertraline Antidepressant Heart Attack Randomized Trial (SADHART), depressed CAD patients randomized to selective serotonin reuptake inhibitor (SSRI) treatment had a numerically lower rate of CVD events than patients randomized to placebo.<sup>22</sup> This suggestive trend was not confirmed in the Myocardial Infarction and Depression Intervention Trial (MIND-IT), in which depressed post-MI patients were randomized to a staged pharmacologic intervention or usual care.<sup>23</sup> Follow-up studies of ENRICHD, SADHART, and MIND-IT confirmed the absence of intervention effects on medical outcomes. 24-26 Interestingly, some post hoc analyses of these trials revealed that patients whose depression improved had better long-term medical outcomes. 24,25,27 However, other researchers have suggested that these relationships may be due to confounding, as early improvements in medical status after a CVD event may predict both later improvements in depressive symptoms and a reduced likelihood of recurrent CVD events. 28,29 This would explain the null intervention effects in these trials.

There are two intriguing exceptions to these negative trials; however, methodological factors cloud interpretation. The first is the TeamCare trial,<sup>30</sup> in which depressed patients with diabetes or CAD were randomized to usual care or blended collaborative care for depression and diabetes/CAD risk factor control. At 12 months, the intervention group exhibited greater improvements in glycated hemoglobin, cholesterol, and blood pressure but not hospitalization rates. Unfortunately, it is unclear whether the depression or diabetes/Revision Date: July 13, 2018

CAD components were responsible for these improvements. The second is the Coronary Psychosocial Evaluation Studies (COPES) trial,<sup>31</sup> in which 6 months of the IMPACT intervention was delivered to persistently depressed CAD patients. At 6 months, intervention patients had fewer CVD events (3 vs. 10), although only 13 total events occurred. Unfortunately, this interesting trend was not maintained in a recent follow-up of this trial.<sup>32</sup> In sum, the critical problem is the absence of interventions to improve CVD outcomes of a large cohort of (depressed) patients at elevated risk of CVD onset, poor CVD prognosis, and high healthcare costs.

A Viable Solution: Treating depression before clinical CVD may yield cardiovascular benefits. Shimbo et al.<sup>33</sup> and others<sup>28,34</sup> have summarized possible reasons for why past depression trials did not detect cardiovascular benefits, including (a) depression differences between treatment and control arms may have been too small to improve CVD outcomes (perhaps due to weak intervention effects, high spontaneous remission rates, or high treatment rates in the control groups), (b) treatment was not initiated while the patient was hospitalized, and (c) the interventions may have been too short (≤6 months). A novel explanation, however, is that the late timing of depression treatment in the natural history of CVD may have played a role. Critically, the past trials all involved patients with preexisting CVD. For several reasons (see b1), we previously hypothesized that treating depression before, versus after, clinical CVD onset could reduce CVD risk.<sup>13</sup>

As a first step, we conducted a follow-up study<sup>35</sup> of Indiana sites of the IMPACT trial,<sup>36</sup> in which older depressed patients were randomized to collaborative care or usual care. We found that IMPACT patients without baseline CVD had a 48% lower risk of a hard CVD event than usual care patients, whereas there was no treatment effect among patients with baseline CVD. Our findings (a) provide preliminary support for our hypothesis that initiating depression treatment before clinical CVD onset may reduce CVD risk and (b) suggest a complement or alternative to the current paradigm of initiating depression treatment after clinical CVD onset to improve CVD prognosis. These unique results strengthen the case that depression is a CVD risk factor and suggest that depression treatment may bring about a clinically relevant reduction in CVD risk.

The IMPACT trial, however, was not designed to test our hypothesis. Consequently, our findings are post hoc and observational, CVD outcomes were not pre-specified endpoints, and virtually no mechanistic data were collected. To address these key limitations, there is a current need for a well-powered, prospective trial.

Establishing that depression treatment reduces CVD risk would have a substantial positive impact. In the scientific domain, a positive trial would vertically advance the field of behavioral medicine in three ways. (1) It would expand the focus of this research area to include delivering depression treatment before, instead of only after, CVD onset. (2) It would remove a critical barrier to progress (past null intervention effects on CVD outcomes) and pave the way for the next step project: a multisite, event-driven Phase 3 trial to confirm elMPACT's efficacy in reducing CVD risk. Specifically, a positive Phase 2 trial would generate the mechanistic rationale (biological plausibility of intervention effects), efficacy evidence (first support of our central hypothesis from a well-powered, prospective trial), and effect size estimates (intervention effects on FMD, candidate mechanisms, and CVD events, which would be combined with estimates from other relevant studies) needed to justify and design a Phase 3 trial. Moreover, a positive Phase 2 trial would further establish the feasibility of our recruitment, intervention, and assessment approaches. (3) The proposed trial will address two long unanswered questions: (a) Is depression a causal risk factor for CVD? (b) What mechanisms underlie the depression-CVD relationship? The lack of experimental evidence, which this trial could generate, prevents depression from being labeled a causal CVD risk factor. In addition, although several plausible mechanisms have been proposed, little direct support has been generated. Elucidating the mechanisms underlying the cardioprotective effect of eIMPACT would allow us to optimize our intervention for CVD risk reduction by adding adjunctive treatments directly targeting the identified mechanisms (e.g., anti-inflammatory medication). In the clinical domain, demonstrating that depression treatment reduces CVD risk, the main expected outcome of this overall line of research, would have a positive impact for three reasons. (1) It would identify a novel target for CVD prevention, likely leading to the inclusion of depression in risk management guidelines. (2) It would equip primary care providers with a new tool (eIMPACT) to simultaneously treat depression and manage the CVD risk of a large cohort of high-risk patients. This tool would also be of use to specialists working with patient groups in which depression is prevalent and CVD risk is high, such as those with diabetes and HIV. 37,38 (3) Positive results, combined our practical intervention, should facilitate the dissemination of eIMPACT. possibly resulting in higher rates of quality depression care. Even though addressing depression in medical settings is a priority, it goes untreated in many patients. Data from a nationally representative sample suggests Revision Date: July 13, 2018

that that only 22% of MDD cases receive adequate care.<sup>3</sup> Demonstrating that a depression intervention reduces CVD risk should move depression treatment up the priority list of both the patient and provider and should encourage healthcare administrators to divert more resources to depression care. In addition, because using a computerized CBT reduces dependence on trained therapists, eIMPACT is more disseminable and scalable, easier to deliver with high fidelity, and likely more cost effective and sustainable than current collaborative care models. Furthermore, eIMPACT has the potential to reach patients with logistical barriers to treatment, such as those in rural areas. eIMPACT's properties (disseminable, scalable, cost-effective, sustainable, and accessible) maximize the public health impact of this line of research.

These three practice changes (identifying a novel treatment target, equipping providers with a new tool, and facilitating intervention dissemination) should reduce CVD morbidity, mortality, and costs, as our preliminary results suggest that treating 1,000 depressed patients may prevent 164 hard CVD events over 5 years.<sup>35</sup> Recently, the American Heart Association set its 2020 Impact Goal, which is "to improve the cardiovascular health of all Americans by 20%, while reducing deaths from CVDs and stroke by 20%." In addition, NHLBI expressed a commitment to reducing socioeconomic status (SES) disparities in CVD in its strategic plan.<sup>39</sup> Given that depression is highly prevalent, especially in low SES groups,<sup>40</sup> depression treatment could play a key role in achieving AHA's goal and in reducing health disparities. Although our preliminary results suggest that a negative trial is unlikely, its importance should not be overlooked. Such an outcome would indicate a need to shift our focus to designing and evaluating alternative approaches to reducing the excess CVD risk of depressed patients (e.g., intervening directly on the underlying mechanisms).

# Innovation

Depression treatment will be delivered before clinical CVD onset, a promising complement or alternative to current paradigm of treating depression in CVD patients to improve CVD outcomes. We propose and report preliminary evidence that treating depression before, versus after, the onset of clinical CVD could yield more pronounced cardiovascular benefits, an idea that is plausible for several reasons.

One, earlier treatment of another CVD risk factor, hypercholesterolemia, produces larger benefits, \$41-43\$ perhaps by slowing atherosclerotic progression. 44 Combining data from trials and prospective studies, Law et al. 42 estimated that the risk reduction in CAD events of a 1.8 mmol/l decrease in LDL cholesterol (achievable with statins) was greater among patients in their 50s (77%) than those in their 60s (61%) and 70s (49%). Other evidence suggests that earlier treatment may slow atherosclerotic progression, as younger age at initiation of statin treatment predicted smaller increases in carotid intima-media thickness over time in children with familial hypercholesterolemia. 44 A recent meta-analysis of genetic studies also bolsters the earlier treatment rationale; it was found that lower LDL cholesterol beginning early in life (due to a mutation) confers a 3 times greater reduction in CAD risk than the same lowering of cholesterol later in life (due to statin treatment). 41 Altogether, these findings raise the possibility that earlier treatment of other modifiable CVD risk factors, including depression, may also slow atherosclerotic progression and prevent CVD events to a greater degree. We are not the first to argue for earlier treatment of CVD risk factors; 45-50 we are just the first to apply this rationale to depression. Steinberg et al. stated that "much of the same reasoning [for hypercholesterolemia] applies to obesity, cigarette smoking, hypertension, diabetes mellitus, and other reversible risk factors" (p. 627). 48

Two, our past work<sup>15,17</sup> and other studies indicate that depression exerts a cardiotoxic influence early in CVD pathogenesis. Depression is reliably associated with endothelial dysfunction<sup>51</sup> and predicts progression of subclinical atherosclerosis in humans<sup>15,17,52,53</sup> and early atherogenesis in primates.<sup>19</sup> Intervening earlier, when depression is exerting a deleterious effect, would minimize exposure to this CVD risk factor.

Three, depression treatments may have greater antidepressive efficacy before clinical CVD onset. Most trials of depressed CVD patients have reported relatively small effect sizes for depression outcomes (0.20-0.38).<sup>54</sup> Similarly, the depressive symptoms effect size observed in our IMPACT follow-up study was 0.06 among depressed patients with baseline CVD; however, it was much larger (0.69) among patients without baseline CVD (see c2.2). A possible explanation is that subgroups of depressed CVD patients in the past trials were experiencing vascular depression<sup>55</sup> (which responds poorly to treatment<sup>56,57</sup>) or an adjustment reaction related to CVD diagnosis and treatment (which is more likely to spontaneously remit<sup>58,59</sup>). Consistent with the latter idea, two trials have reported medium effect sizes in CVD patients with persistently elevated depressive Revision Date: July 13, 2018

symptoms.<sup>31,60</sup> Because we will enroll depressed patients without clinical CVD, our sample should have few patients from the subgroups thought to be contributing to the smaller effect sizes of past trials.

Four, conventional prognostic factors, such as CVD event severity or cardiovascular interventions (e.g., revascularization procedures), may override the effect of depression during the later stages. 16,61

We will examine multiple candidate mechanisms of elMPACT's hypothesized effect on CVD risk. As we have done previously, <sup>15</sup> we will conduct formal statistical mediation tests to examine the leading candidate mechanisms through which depression treatment may reduce CVD risk – i.e., decreases in depressive symptoms, autonomic dysfunction, systemic inflammation, and platelet activation. We will also explore atherogenic behavioral factors, conventional CVD risk factors, and depression care variables as potential mechanisms (see c3.5). Although many plausible mechanisms have been proposed previously, testing for mediation is rare in this field, <sup>62</sup> particularly in the favorable context of a RCT, which allows for stronger inferences. The proposed study would be the first prospective trial to examine candidate mechanisms underlying the hypothesized cardioprotective effect of depression treatment initiated before CVD onset.

# elMPACT is a novel intervention and an appropriate selection for the proposed trial.

Although collaborative depression care has been examined in CVD patients, <sup>31,60,63</sup> no trials in this area have incorporated computerized psychotherapy into this framework. The original IMPACT intervention is an established, collaborative, stepped care program involving a multidisciplinary team delivering evidenced-based treatments (antidepressants and psychotherapy) consistent with patient preference. <sup>36,64,65</sup> We will modernize the IMPACT intervention (a) by adding a computerized CBT, Beating the Blues (BtB), as the first-line psychotherapy and (b) by delivering other components, including Problem Solving Treatment in Primary Care (PST-PC), via telephone. BtB is a stand-alone CBT program for depression designed for primary care patients and appropriate for adults with lower reading levels and computer experience. <sup>66</sup> BtB uses an interactive, multimedia format to deliver 8 weekly sessions, the structure and content of which mirror face-to-face CBT. We will also deliver PST-PC via telephone, which Davidson et al. <sup>60</sup> recently found to be feasible and efficacious.

In addition to being novel, there are two reasons why eIMPACT is an appropriate selection. First, the eIMPACT components are efficacious and acceptable. In the IMPACT trial, <sup>36</sup> 45% of intervention patients versus 19% of usual care patients had >50% reduction in depressive symptoms, and satisfaction was high. In our IMPACT follow-up study, <sup>35</sup> we observed a moderate to large effect size for depressive symptoms (see c2.1). BtB has more empirical support than any other computerized psychotherapy, including a positive RCT of 274 primary care patients. <sup>67,68</sup> BtB has been found to be a potent intervention, <sup>67-75</sup> with effect sizes comparable to face-to-face CBT. <sup>76</sup> In our pilot trial, we observed a large BtB effect size for depressive symptoms (see c2.2). BtB has been shown to be acceptable to patients <sup>66,74,75</sup> and was recently found to be effective, acceptable, and preferred to usual care among older adults. <sup>77</sup> In 2006, NICE recommended BtB for managing depression in the English National Health Service. <sup>78</sup> Early studies in the U.S. are promising, <sup>79</sup> and large trials are underway (including Dr. Rollman's trial; NCT01482806). Because we are retaining the key elements of the IMPACT model and our pilot data support the efficacy of BtB in the target population, we expect eIMPACT to achieve an effect size as large as the original IMPACT intervention with fewer human resources.

Second, eIMPACT fits very well with our long-term goal of developing, optimizing, and disseminating treatments to improve the CVD outcomes of a large cohort of patients at elevated risk of CVD onset, poor CVD prognosis, and high healthcare costs. To achieve this goal, large-scale dissemination and adoption must be possible. Because eIMPACT uses a stand-alone computerized CBT, it is more disseminable and scalable, easier to deliver with high fidelity, and likely more cost effective<sup>80</sup> and sustainable than current collaborative care models. Given that components of eIMPACT are computer and telephone delivered, it also has the potential to reach patients with logistical barriers. Finally, implementation tools for the IMPACT intervention are available (see <a href="impact-uw.org">impact-uw.org</a>) and could be leveraged to facilitate dissemination and adoption of eIMPACT.

Our trial design is not ideal for determining the differential efficacy of the eIMPACT components. If that was our goal, we would have chosen a 2 Antidepressants (yes, no) x 2 CBT (yes, no) design. While such a study would be valuable, our trial is the preferable next step in our view. First, we selected a flexible and efficacious treatment model to achieve our broader objective of determining whether successfully treating depression earlier in the natural history of CVD reduces CVD risk. Second, dismantling eIMPACT could neutralize some Revision Date: July 13, 2018

key strengths (i.e., stepped care, patient choice, and treat to target), potentially compromising its efficacy. Third, justifying the higher cost of a dismantling study is difficult when the intact treatment has not been shown to reduce CVD risk in a prospective trial. Based on our IMPACT follow-up study,<sup>35</sup> we expect eIMPACT patients to receive both antidepressants and CBT (50%), antidepressants only (26%), CBT only (12%), or neither component (12%). To generate hypotheses, we propose supplemental analyses to explore which components are most strongly related to the outcomes (see c3.5).

# Brachial flow-mediated dilation (FMD) is an innovative and appropriate primary outcome.

The proposed trial would be the first to examine the effect of depression treatment, delivered before clinical CVD onset, on endothelial dysfunction. Endothelial dysfunction, the impaired ability of the vascular lining to maintain normal homeostasis, <sup>81</sup> is an early precursor to and plays a central role in atherosclerosis. <sup>82</sup> FMD is a noninvasive technique that uses high-resolution ultrasound to measure changes in brachial diameter in response to stimuli, <sup>83</sup> with results correlating closely with coronary endothelial function. <sup>84,85</sup> Measurements are made before and after endothelium-dependent and endothelium-independent stimuli. <sup>86</sup> The endothelium-dependent stimulus is hyperemic blood flow triggered after the release of an inflated blood pressure cuff around the forearm. The shear stress from the increased blood flow causes endogenous vasodilators (e.g., nitric oxide) to be released from the endothelium, which relaxes the vascular smooth muscle. This dilation of the brachial artery is thus a measure of the endothelium's ability to respond normally to hyperemic shear stress. Nitroglycerin, the endothelium-independent stimulus that directly relaxes smooth muscle, is then applied to assess the smooth muscle's functional capacity. If FMD is low and nitroglycerin-mediated dilation is normal, the endothelium (and not the smooth muscle) can be safely assumed to be dysfunctional.

FMD is the best choice for the primary outcome of the proposed trial for several reasons. One, endothelial dysfunction is considered a barometer of total CVD risk and the final common pathway through which CVD risk factors promote atherosclerosis. 87-89 Endothelial dysfunction (a) has been observed in adults with CVD risk factors but no detectable disease, 83,90-97 (b) is related to other vascular disease measures, 98-100 and (c) is an independent predictor of CVD events among initially healthy persons, at-risk individuals, and CVD patients. 101-<sup>112</sup> Two, intervention-related improvements in FMD predict a reduced incidence of CVD events, <sup>113-115</sup> indicating that FMD is a predictor of clinical benefit. In contrast to anatomic measures such as coronary calcification and carotid thickness, FMD also responds within weeks of pharmacologic and behavioral interventions.<sup>87</sup> making it well suited to evaluate if a new treatment approach holds promise. Three, FMD is a continuous measure of CVD risk that provides greater statistical power than dichotomous outcomes. Thus, trials with FMD as the primary outcome require much smaller samples and shorter follow-ups than CVD event-driven trials. Four, a recent meta-analysis<sup>51</sup> and our pilot findings (see c2.3) demonstrate that depressed adults exhibit evidence of endothelial dysfunction as measured by FMD relative to their nondepressed counterparts. Although results of some surrogate endpoint trials have not been confirmed in subsequent event-driven trials, 116 this risk is minimized here. First, we have already detected a beneficial effect of a similar intervention on CVD events in our post hoc analysis of the IMPACT trial, 35 increasing the likelihood that we will see a comparable effect in a prospective, event-driven Phase 3 trial. Second, in the proposed Phase 2 trial, we will collect event data and explore whether eIMPACT patients show a clinically relevant reduction in events.

# Using a statewide information exchange to identify CVD events is unique and has advantages.

We will leverage this unique resource to identify CVD events. The Indiana Network for Patient Care (INPC), 117,118 the nation's largest clinical data repository (see Facilities and Other Resources), was an NIH-funded expansion of the Regenstrief Medical Record System, 119 which has been used extensively for clinical research. The INPC contains 4.7 billion bits of standardized clinical data for 14.7 million patients from 19,000 physicians, 90 hospitals, and 110 clinics and other sites. The participating systems deliver registration records; coded diagnoses and procedures; laboratory, pathology, and vital signs data; emergency department, inpatient, and outpatient encounter data; and pharmacy data. INPC also gathers data from Indiana Medicaid and other commercial payers, as well as death data from the Indiana State Department of Health.

Advantages of our approach include minimal attrition and an observation period that can be easily extended. As in our IMPACT follow-up study,<sup>35</sup> we anticipate having event data for nearly all randomized patients, given that (a) we will identify most CVD events through INPC searches (no patient participation required) and (b) we have developed procedures (e.g., follow-up calls) to identify the few events that may occur outside of the INPC

catchment area. Extending the observation period to capture more CVD events would also require few resources, as it would involve the data manager re-running INPC search programs.

# **Proposed Research and Conceptual Framework**

We will conduct a Phase 2 randomized controlled trial of 220 primary care patients aged 50+ years with a depressive disorder and CVD risk factors but no clinical CVD. Patients will be randomized to 12 months of eIMPACT or usual care and will be followed for a mean of 4 years. The conceptual framework guiding our trial is shown in Figure 1. Our central hypothesis is that eIMPACT will improve endothelial dysfunction by decreasing depressive symptoms, autonomic dysfunction, systemic inflammation, and platelet activation.

The atherogenic physiologic and behavioral factors in Figure 1 are the leading candidate mechanisms through which depression treatment may reduce CVD risk. Substantial literatures indicate that depression is reliably associated with each factor, 120-126 as well as endothelial dysfunction. Although far fewer in number, some studies have reported more direct evidence. We and others have observed that the strength of the depression-CVD association is attenuated after adjusting for autonomic function indices, 127,128 inflammatory markers, 128-130 physical activity, 130-133 and smoking. 15,130,131,133 Finally, evidence suggests that CBT and SSRIs decrease autonomic dysfunction, 134-137 inflammation, 138-143 platelet activation, 144-147 and smoking. While we propose that treatment-related reductions in depressive symptoms (paths a and b) will result in decreases in the atherogenic factors (paths d and e), we also hypothesize that SSRIs and SNRIs will reduce CVD risk via their

Figure 1. Conceptual Framework of the Proposed Clinical Trial



direct effects on inflammation and platelet activation (path c). <sup>33,147,150</sup> We chose the physiologic factors as secondary outcomes, given that they represent likely pathways through which behavioral factors increase CVD risk (path f). This conceptualization is in line with current models of the depression-CVD relationship<sup>151</sup> and empirical findings. <sup>152-155</sup> We will examine behavioral factors as mechanisms in exploratory analyses.

2.0 Rationale and Specific Aims

Cardiovascular disease (CVD) is a top public health concern in the U.S. CVD is highly prevalent and is the number one killer of Americans. Moreover, its economic burden is substantial and on the rise. 1,2 Thirty years of evidence indicates that adults with depression are at increased risk of CVD events and poor CVD prognosis; 8,9 however, attempts to improve the CVD outcomes of depressed patients have been unsuccessful. The few trials 21-23,30-32 that have evaluated whether depression interventions reduce the likelihood of CVD events generally have not observed the anticipated benefits. The reasons for these null results have been the subject of debate. 34 We recently proposed a novel explanation: the depression interventions in these trials, all of which involved patients with preexisting CVD, may have been delivered too late in the natural history of CVD. 13 We hypothesized that treating depression before, versus after, the onset of clinical CVD could reduce CVD risk because: (1) earlier treatment of another CVD risk factor, hypercholesterolemia, yields more pronounced benefits, 41-44 (2) depression exerts a cardiotoxic influence early in CVD pathogenesis, 17,19,51,53 (3) depression treatments appear to have greater antidepressive efficacy prior to clinical CVD onset, 36,54 and (4) conventional prognostic factors may override depression's harmful effect during the later stages of CVD.

As a first step, we conducted an 8-year follow-up study<sup>35</sup> of Indiana sites of the Improving Mood-Promoting Access to Collaborative Treatment (IMPACT) trial,<sup>36</sup> in which older depressed patients were randomized to a collaborative care intervention or usual care. Results supported our hypothesis. Intervention patients without baseline CVD had a 48% lower risk of myocardial infarction (MI) or stroke than usual care patients. There was no treatment effect among patients with baseline CVD. Although these results are unique and potentially significant, the IMPACT trial was not designed to test our hypothesis. Thus, our findings are post hoc and observational, CVD outcomes were not pre-specified endpoints, and virtually no mechanistic data were collected. To address these key limitations, there is a current need for a well-powered, prospective trial. Revision Date: July 13, 2018

Our long-term goal is to develop, optimize, and disseminate treatments to improve CVD outcomes of a large cohort of patients at elevated risk of CVD onset, poor CVD prognosis, and high healthcare costs. This project's objective is to test whether our modernized IMPACT intervention (eIMPACT), delivered before CVD onset, reduces CVD risk. We propose a Phase 2 randomized controlled trial of 220 primary care patients (≥50 years, 40% African American) with a depressive disorder and CVD risk factors but no clinical CVD. Patients will be randomized to 12 months of eIMPACT (a collaborative stepped care program including antidepressants and computerized and telephonic cognitive-behavioral therapy) or usual care (usual primary care for depression). Patients will be followed for a mean of 4 years. The primary outcome is endothelial dysfunction assessed by brachial flow-mediated dilation (FMD),<sup>81</sup> which is considered a barometer of CVD risk.<sup>88</sup> Critically, intervention-related improvements in FMD predict a reduced incidence of CVD events.<sup>113-115</sup> Our central hypothesis is that eIMPACT will improve endothelial dysfunction in depressed patients by decreasing depressive symptoms, autonomic dysfunction, systemic inflammation, and platelet activation, which are leading candidate mechanisms. We will test our central hypothesis by carrying out these specific aims:

Aim 1: Determine whether elMPACT reduces the excess CVD risk of depressed patients. Depressed patients randomized to elMPACT, versus usual care, will exhibit a clinically and statistically significant improvement in the primary outcome of endothelial dysfunction at the 12-month post-treatment visit (Hypothesis 1). We will also explore whether elMPACT patients, versus usual care patients, show a clinically relevant reduction (25% lower relative risk<sup>156,157</sup>) in CVD events (exploratory outcome) over a mean observation period of 4 years (1-year intervention period plus 3-year follow-up period).

Aim 2: Examine candidate mechanisms underlying the effect of elMPACT on CVD risk. Depressed patients randomized to elMPACT, versus usual care, will exhibit greater decreases in the secondary outcomes of depressive symptoms (Hypothesis 2), autonomic dysfunction (Hypothesis 3), systemic inflammation (Hypothesis 4), and platelet activation (Hypothesis 5) at the 12-month post-treatment visit. We will also explore whether decreases in these four candidate mechanisms (a) are associated with improvements in endothelial dysfunction and (b) are partial mediators of elMPACT's hypothesized cardioprotective effect.

A positive trial would generate the mechanistic rationale, efficacy evidence, and effect size estimates needed to justify and design a multisite, event-driven Phase 3 trial to confirm elMPACT's efficacy in reducing CVD risk. Conversely, a negative trial would indicate a need to evaluate alternative approaches to reducing the excess CVD risk of depressed patients. Demonstrating that depression treatment reduces CVD risk, the main expected outcome of this line of research, would have a substantial positive impact. It would identify a novel target (depression) for CVD prevention efforts, and it would equip providers with a new disseminable and scalable tool (elMPACT) to treat depression and manage the CVD risk of a large cohort of high-risk patients. These clinical practice changes should translate into reduced CVD morbidity, mortality, and costs, as our preliminary results suggest that treating 1,000 depressed adults may prevent 164 CVD events over 5 years. 

\*\*These clinical practice changes should translate into reduced CVD morbidity, mortality, and costs, as our preliminary results suggest that treating 1,000 depressed adults may prevent 164 CVD events over 5 years.

### 3.0 Inclusion/Exclusion Criteria

# Inclusion criteria

- Primary care patients
- Age ≥ 50 years
- Current depressive disorder
- Elevated CVD risk

To identify patients with a current depressive disorder, ResNet assistants will administer the PHQ-9, $^{158}$  a validated diagnostic measure designed for primary care patients. $^{159-162}$  We will consider patients to have a depressive disorder if (a) they have a PHQ-9  $\geq$ 10 $^{158}$  and (b) they meet criteria for a PHQ-9 depressive disorder diagnosis (2 or more of the 9 depressive symptoms, including depressed mood or anhedonia, present in the past two weeks). $^{160}$  The cut point of  $\geq$ 10 has 88% sensitivity and 88% specificity for MDD diagnosed by a clinical interview. $^{158}$  The combination of a PHQ-9  $\geq$ 10 and a PHQ-9 depressive disorder diagnosis helps to ensure that false positives will not be enrolled. In addition to its diagnostic validity, we chose a PHQ-9 case finding approach because: (a) it is feasible in primary care and is how depressed patients will likely be

identified in clinical practice, (b) recent successful trials have used similar approaches, <sup>31,60,163</sup> and (c) we observed evidence of a signal of depression treatment on endothelial function and inflammation in our pilot trial, in which we used the PHQ-9.

Elevated CVD risk will be defined as  $\geq 1$  (if 60+ years) or  $\geq 2$  (if 50-59 years) of the following risk factors in the medical record in the past 5 years but no clinical CVD: hypertension, hypercholesterolemia, diabetes, or current smoking. According to the Framingham risk calculator for primary care patients, <sup>164</sup> the odds of a CVD event of a 50-year-old man/woman with 2 risk factors is about equivalent to that of a 60-year-old man/woman with 1 risk factor.

### **Exclusion Criteria**

- History of clinical cardiovascular disease
- Presence of the following chronic disorders: HIV/AIDS, chronic kidney disease, or active cancer/current cancer treatment
- History of bipolar disorder or psychosis
- Continuous (e.g., daily) treatment for a systemic inflammatory condition (e.g., rheumatoid arthritis, lupus, Crohn's disease, and ulcerative colitis) in the past 3 months. Nonsteroidal anti-inflammatory drug (NSAID) use is allowed, given its high prevalence in the target population.
- Current use of anticoagulants (Aspirin and cholesterol and blood pressure medications are allowed.)
- Acute risk of suicide
- Severe cognitive impairment (≥3 errors on 6-item cognitive screen<sup>165</sup>)
- Current pregnancy
- Ongoing depression treatment with a psychiatrist outside of the Eskenazi Health/Midtown system (ongoing depression treatment with a Eskenazi Health/Midtown psychiatrist is allowed, as we will be able to collaborate and coordinate depression care)

A history of clinical CVD will be defined as any of the following in the medical record before enrollment: CAD (ICD-9 410-414, 429.2) or CBV (ICD-9 430-434) diagnosis, acute MI (CK-MB >3.0 ng/ml or troponin >0.3 μg/L), percutaneous coronary intervention (ICD-9 00.66, 36.03, 36.06, 36.07, 36.09; CPT 92980-92984, 92995, 92996), or coronary artery bypass graft (ICD-9 36.10-36.19; CPT 33510-33536).

#### 4.0 Enrollment/Randomization

We will use the 3-stage process of our past trials to recruit patients. First, the Regenstrief Medical Records System, one of most comprehensive electronic medical records, will be searched in accordance with HIPAA to generate lists of eligible patients. Next, ResNet assistants will obtain permission to approach from each patient's provider. ResNet, Indiana University's primary care practice-based research network, is the sole mechanism through which patients in the targeted clinics can be contacted for research. ResNet also maintains a patient registry, which will also be used by ResNet to identify potentially eligible patients. Finally, ResNet assistants will conduct high-intensity in-clinic and telephone screening and will enroll eligible patients (see Appendix 1 for Screening Interview). ResNet assistants will use a paper copy or a REDCap version of the Screening Interview. Through administering the eligibility interview refined in our pilots, ResNet assistants will assess cognitive function, medical/psychiatric status, and depression status; will obtain consent and authorization; and will implement the suicidal ideation protection protocol.

We estimate that ≈4,320 patients (45/week) will need to be approached, consistent with the IMPACT trial.<sup>36</sup> We will be able to start recruitment immediately, as the infrastructure, personnel, and protocols are in place from the PI's recent trials. At the Indiana sites of the IMPACT trial, 6.4% of approached patients were randomized. We conservatively estimate that 5% of approached patients will be randomized (9/month) in the proposed trial. Patients who meet inclusion/exclusion criteria and consent will be scheduled for the pre-treatment visit. Because only patients who attend this visit will be randomized, it will serve as a prerandomization compliance screening.<sup>167</sup>

In the unanticipated event of slower-than-projected recruitment, we will first request direct referrals from providers in the targeted clinics. Next, we will pursue expanding recruitment to another healthcare system in Indianapolis, such as the VAMC or Community Health Network. Finally, we will extend the recruitment window up to a year if the benefits to the primary outcome of endothelial dysfunction (ample power due to a larger sample) outweigh the costs to the exploratory outcome of CVD events (shorter observation period).

At the end of the pre-treatment visit described below, the randomization procedure will be initiated. To balance the groups on two strong FMD correlates,<sup>91</sup> randomization will be stratified by sex and age (50-59 and 60+ years) using random number sequences.<sup>168</sup> Sequentially numbered sealed envelopes containing group assignment will be prepared by the study statistician (Dr. Gao).

# 5.0 Study Procedures

### Overview, Visits, and Setting

We will conduct a Phase 2 randomized controlled trial of 220 primary care patients aged 50+ years with a depressive disorder and CVD risk factors but no clinical CVD. Patients will be randomized to 12 months of eIMPACT, our modernized IMPACT intervention, or usual care and will be followed for a mean of 4 years.

The timing of activities is shown in the table below. We will strive to schedule patients within two weeks of enrollment, although some visits will fall outside of that window due to conflicts in the patients' schedules and no-showed or rescheduled appointments. Patients will attend a 3-hour pre-treatment visit at the Indiana CTSI Clinical Research Center. To minimize the effect of extraneous factors on FMD, 169,170 patients will be told to fast and to avoid tobacco and exercise for ≥8 hours before their visit. The exam room will be kept at 68-71°F, and premenopausal women will be scheduled within 2 weeks of menstruation onset. Patients will have their height, weight, and BP measured; will complete self-report scales on a secure SurveyMonkey website designed for this study visit; and will undergo FMD and heart rate variability assessments and a blood draw (standard venipuncture). To end this visit, the randomization procedure will be initiated, the patient and the treatment team will be notified of the assignment, and the mid-treatment call and post-treatment visit will be scheduled. If the patient is randomized to the eIMPACT intervention, the depression clinical specialist will conduct a brief session over FaceTime to orient the patient to intervention materials and to schedule the initial assessment. The FaceTime session will not be recorded. Within 2 weeks, the depression clinical specialist will call eIMPACT patients to initiate treatment, and a research assistant will send a letter to the primary care providers of usual care patients to notify them that their patient has a depressive disorder and to encourage follow-up. Approximately six months after randomization, research assistants will contact all patients to complete the 45-min mid-treatment call. First, a brief questionnaire used in our pilot trials will be administered to assess for the occurrence of CVD events since enrollment. As we have also done in our pilot projects, the self-reported scales completed at pre-treatment will then be readministered. Approximately twelve months after randomization, patients will return to the Clinical Research Center for the post-treatment visit, during which all factors measured at pre-treatment will be reassessed. Finally, research assistant will contact patients annually after their post-treatment visit to complete the follow-up calls, with the last call coming within 2 weeks of the study end date. These calls will follow the same procedures as the mid-treatment call.

The schedule of participant reimbursement is as follows: \$100 for the pre-treatment visit, \$25 for the mid-treatment call, \$100 for the post-treatment visit, \$20 for each of the annual follow-up calls, and up to \$10 per visit to cover parking or transportation costs.

| | Υ | ear 0 | 1 | Υ | 'ear 0 | 2 | Υ | ear 0' | 13 | Υ | 'ear 0 | 4 | Υ | ear C | 5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Recruitment & Pre-Treatment Visits | | | | | | | | | | | | | | | |
| Treatment | | | | | | | | | | | | | | | |
| Mid-Treatment Calls | | | | | | | | | | | | | | | |
| Post-Treatment Visits | | | | | | | | | | | | | | | |
| Annual Follow-Up Calls | | | | | | | | | | | | | | | |
| Analysis & Manuscript Submission | | | | | | | | | | | | | | | |

The setting, which is identical to the IMPACT trial, is the primary care clinics of two healthcare systems affiliated with Indiana University: Eskenazi Health and Indiana University Health. Eskenazi Health, a safety net

healthcare system, provides care for ≈20% of the population of Indianapolis. The Eskenazi Health Center for Senior Health, where elderly patients receive primary care, is included in the targeted clinics. About 90% of Eskenazi patients are underinsured or uninsured, and 50% are African American. Therefore, these patients provide special opportunities to research diseases that disproportionately affect lower SES and minority populations, such as CVD.<sup>1,171</sup> Indiana University Health, a large academic medical center, is Indiana's most comprehensive healthcare system.

# **Treatment Groups**

#### *eIMPACT*

eIMPACT is a collaborative stepped care intervention involving a multidisciplinary team delivering evidenced-based treatments consistent with patient preference. We will modernize the IMPACT intervention (a) by adding a computerized CBT as the first-line psychotherapy and (b) by delivering some of the other components via telephone or FaceTime (see below). None of the computerized, telephonic, or FaceTime sessions will be recorded. Other than restricting the list of antidepressant medications to maximize CVD risk reduction, the remaining IMPACT components will not be altered.

Beating the Blues (BtB; Ultrasis PLC) is a widely used, empirically supported, stand-alone CBT program for depression designed for primary care patients and appropriate for adults with little computer experience and a 5<sup>th</sup>-6<sup>th</sup> grade reading level.<sup>66</sup> In prior trials, we have used the UK and US versions; we will use the US version in the proposed trial (see <a href="www.beatingthebluesus.com">www.beatingthebluesus.com</a> for a brief video tutorial). BtB utilizes an interactive, multimedia format to deliver eight 50-minute, weekly sessions, the structure and content of which mirror face-to-face CBT. Although sessions are tailored to each patient's problems, general topics include challenging dysfunctional thoughts, activity scheduling, problem solving, graded exposure, task breakdown, sleep management, and relapse prevention. Patients are also assigned tailored homeworks.

To minimize treatment barriers (e.g., transportation issues) and attrition, to reduce subject burden, and to ultimately facilitate implementation of eIMPACT, BtB sessions will occur in a private room at the Clinical Research Center, at Dr. Stewart's laboratory, at the patient's primary care clinic, or in a location selected by the patient where s/he can access a computer with internet, such as the patient's home, the patient's work, a family member's/friend's home, or a public library. Patient preference will drive the location decision. Patients will be offered with ear bud headphones if they plan to use them at remote locations and do not already own a pair that they would rather use. All patients completing BtB will be provided with a BtB binder that contains printouts of all BtB worksheets.

To begin each in-person BtB session, an assistant will collect the homework. The patient will then work alone through the BtB session at his/her own pace, with the assistant providing help only with technical issues. To end the session, the assistant will give the patient the printed homework.

Remote BtB sessions will scheduled, just like in-person sessions. To begin each remote BtB session, an assistant call the patient to instruct the patient to put last week's homework in the BtB binder, to address any technical issues, and to ensure that the patient has launched the correct BtB session for that day. The patient will then work alone through the BtB session at his/her own pace, with the assistant monitoring progress remotely on the secure BtB website set up for this trial. To end the session, the assistant will call the patient back to address any questions and ensure that the patient has identified the correct printed homework in the BtB binder.

Problem Solving Treatment in Primary Care (PST-PC) is a manualized, empirically supported CBT developed for use by healthcare professionals in primary care. The focus of the 6-10 30-minute sessions is teaching patients approaches for solving current problems contributing to depression. PST-PC was the first-line therapy in the IMPACT trial; however, it is our second-line therapy. We will deliver PST-PC primarily via telephone or FaceTime (although in-person sessions are also allowed), which Davidson et al. fo found to be feasible and efficacious in the recent CODIACS Vanguard trial. Our consultant (Dr. Rollman) also completed the Bypassing the Blues trial in which his team delivered collaborative depression care to cardiac patients via telephone and observed positive results.

The IMPACT treatment manual provides guidelines for using antidepressants, such as selecting a medication, titrating, switching to another medication, managing side effects, and avoiding drug interactions. <sup>65</sup> To optimize eIMPACT for CVD risk reduction, we have restricted the IMPACT list of antidepressants to SSRIs, duloxetine, bupropion, and mirtazapine. These medications are FDA approved for the treatment of depression and are the safest from a cardiovascular perspective. <sup>178,179</sup> We are prohibiting the use of most serotonin-norepinephrine reuptake inhibitors (SNRIs) and all tricyclics due to their potential adverse effects on cardiovascular parameters. <sup>178,179</sup> We do not expect this change to have a negative effect on depression outcomes, as antidepressants not on our list of allowed medications are typically used only as second- or third-line treatments and also have contraindications. <sup>65</sup>

At the first session, the depression clinical specialist (DCS), a Master's-level licensed mental health counselor (LMHC), will review depression materials and discuss treatment options. The DCS will then work with the patient's primary care provider to develop a plan that follows the IMPACT algorithm<sup>65</sup> with modifications noted above. Our modernized algorithm recommends a Step 1 treatment of 8-12 weeks of BtB or an antidepressant depending on the patient preference. Providers will manage prescriptions. In addition to delivering PST-PC, the DCS will help the patient adhere to antidepressant therapy and schedule pleasurable activities. If the patient is taking an antidepressant at baseline, the dose will be increased, BtB will be added, or the antidepressant will be discontinued and another one will be prescribed or BtB will be delivered. If the patient wants psychotherapy but has a strong preference for traditional treatment, PST-PC will be offered at Step 1. The DCS will have weekly team meetings with the supervising psychiatrist (Dr. Nurnberger) and primary care expert (Dr. Callahan), during which new cases and those requiring plan changes will be discussed. Fidelity to the eIMPACT algorithm will be continually assessed and recorded by the supervisors at these team meetings, and adjustments needed to ensure high fidelity will be made.

The DCS will follow patients for 12 months, while monitoring response. <sup>158</sup> At the start, the DCS will attempt to have telephone sessions or contacts at least every 2 weeks. For patients who achieve remission (≥50% PHQ-9 reduction and <3 MDD symptoms<sup>36</sup>), the DCS will develop a relapse prevention plan and follow up monthly. Step 2 treatment – which involves either augmenting Step 1 treatment with an antidepressant or psychotherapy or switching to another antidepressant or psychotherapy – will be delivered to patients who do not achieve remission. If a patient does not respond after 6-10 more weeks, Step 3 treatment will be initiated, which consists of additional medications and psychotherapy, hospitalization, or other services. In the IMPACT trial, <sup>36</sup> intervention patients had 9.2 ± 6.2 in-clinic sessions and 6.1 ± 5.1 telephone contacts with a DCS during the 12 months of treatment. At the end of the 12 month treatment phase, the participant will receive a certificate indicating completion of elMPACT treatment. We expect similar numbers in our trial, although most sessions/contacts will be via telephone. Based on our experiences, one DCS can manage 80-100 patients. The maximum number of patients in treatment at any given time in this trial will not exceed 80.

#### **Usual Care**

This arm was modeled after the IMPACT trial control group. 36 At the pre-treatment visit, patients will be informed of their depression diagnosis and group assignment, will be provided with a list of local mental health services (with contact information) available to Eskenazi patients, and will be encouraged to follow-up with their primary care provider regarding their depression. These patients will also be reminded (from the informed consent statement) that, although we will pass along information to their primary care provider, participants in this group do not receive any depression treatment from the study team; instead, all depression treatments that participants in this group receive during the study are delivered by their usual providers. The patient's PCP will also receive a letter indicating that their patient has a depressive disorder and was randomized to usual care. This letter will encourage the PCP to follow-up with their patient to address their depression, will note that there are no restrictions on the care that these patients can receive, and will provide the same list of Eskenazi mental health services given to patients. Although this feedback could result in treatment that would not have occurred naturally in primary care, informational support alone is unlikely to improve depression outcomes. 180 Moreover, our pilot trial indicates that depression outcomes achieved with usual care in targeted clinics remain suboptimal (see c2.2). Patients in both arms will continue to have access to services that are part of usual care in the targeted systems. There will be no restrictions on the care received, although new depression treatments received outside of the trial are discouraged in the eIMPACT group.

<u>Assessments</u>

| | Pre-Treatment*<br>(0 months) | Mid-Treatment <sup>†</sup><br>(6 months) | Post-Treatment*<br>(12 months) | Annual Calls†<br>(2-4 calls) |
|---|---|---|---|---|
| Endothelial Dysfunction (Primary Outcome) | X | | X | |
| Atherogenic Physiologic Factors (Secondary Outcomes) | X | | X | |
| Depressive Symptoms (Secondary Outcome) | X | X | X | X |
| CVD Events (Exploratory Outcome) | | X | X | X |
| Atherogenic Behavioral Factors | X | X | X | X |
| Conventional CVD Risk Factors | X | | X | |
| Miscellaneous Factors | X | X | X | X |

<sup>\*</sup>Clinical Research Center Visit. †Telephone Call.

### Endothelial Dysfunction (Primary Outcome)

Patients will undergo FMD assessments at Dr. Gupta's laboratory in accordance with consensus guidelines.<sup>81</sup> Dr. Gupta as well as Ms. Grounds and Ms. Scott (our vascular ultrasonographers) have undergone certified training through the University of Wisconsin Brachial Artery Reactivity Testing Symposium. Our group has performed 700+ FMD assessments in the past 10 years. We utilize a GE Logiq E ultrasound system with AccessPoint 2011 software. To illustrate the reproducibility of our results, we performed paired FMDs over 1-4 weeks in 11 healthy volunteers in 2013. Intraclass correlations for baseline diameter, reactive hyperemia, and FMD were 0.98, 0.98, and 0.70, which compare favorably to other laboratories.<sup>181-183</sup>

After a 10-minute supine rest, high-resolution baseline images of the brachial artery will be obtained from 3 consecutive cardiac cycles. Next, the forearm cuff will be inflated to 250 mmHg for 5 minutes and then rapidly deflated. At 60 and 90 seconds post deflation, images from 3 consecutive cardiac cycles will be acquired. Brachial diameters will be measured at peak R wave. FMD values will be computed as % increase in diameter at 60 or 90 seconds post deflation<sup>196,197</sup> (the larger of the two values). Percent change in reactive hyperemic flow velocities will also be computed to ensure that sufficient shear stress triggers were induced.

### Atherogenic Physiologic Factors (Secondary Outcomes)

To quantify autonomic function, we will assess high-frequency heart rate variability, a parasympathetic index, following established guidelines. <sup>184,185</sup> See our paper <sup>186</sup> for complete details. Briefly, using an electrode arrangement recommended by Qu et al., <sup>187</sup> a HIC-2000 impedance cardiograph, and MindWare software, estimates of high-frequency heart rate variability (In of ms²/Hz) will be derived by spectral analysis (bandwidth: 0.15-0.40 Hz) from 1-minute epochs of ECG data obtained during the last 5 minutes of a 10-minute rest period. To control for the influence of respiration rate on high-frequency heart rate variability, participants will complete a paced-breathing computer task set to a normal resting rate of 12 breaths/minute during ECG data collection. Values will be corrected for respiration. <sup>188,189</sup> Blood samples obtained by research nurses from the median cubital vein will be centrifuged within 20 minutes. Plasma aliquots will be frozen at -80°C until the time of assay at the Indiana CTSI Clinical Research Assay Laboratory directed by Dr. Considine. To quantify systemic inflammation, we will measure IL-6 and CRP levels using R&D Systems ELISA kits. To quantify platelet activation, we will measure levels of platelet-specific release products, β-thromboglobulin (BTG) and platelet factor 4 (PF4), <sup>190</sup> using R&D Systems ELISA kits. The remaining plasma aliquots will saved for possible future assays. Assistants scoring the autonomic data and performing the assays will be blind to assignment.

### Depressive Symptoms (Secondary Outcome)

Like the IMPACT trial,<sup>36</sup> we will assess depressive symptoms with 20 depression items of the Symptom Checklist-90 (SCL-20), a reliable and valid measure.<sup>191-194</sup> We will examine total score and % remitted. We also added an item ("Sleeping too much") to the SCL-20 to measure this symptom of atypical depression that was not including in the original questionnaire. We will also administer the PHQ-9 to assess depressive symptoms.

# CVD Events (Exploratory Outcome)

Our exploratory outcome, modeled after the JUPITER trial, <sup>195</sup> is time to first major CVD event, defined as: <u>CVD death</u> (ICD-10 I20-I25 or I60-I69 the first-listed cause of death); <u>nonfatal MI</u> (CK-MB >3.0 ng/ml, troponin >0.3 µg/L, or ICD-9 410); <u>nonfatal stroke</u> (ICD-9 430-432, 433.01, 433.11, 433.21, 433.31, 433.91, 434.01, 434.11, 434.91); <u>unstable angina</u> requiring hospitalization (inpatient admission ICD-9 411.1); and <u>revascularization</u> – i.e., percutaneous coronary intervention (ICD-9 00.66, 36.03, 36.06, 36.07, 36.09; CPT 92980-92984, 92995, 92996) or coronary artery bypass graft (ICD-9 36.10-36.19; CPT 33510-33536). Because recruitment will occur during Years 01-02, the mean observation period will be 4 years (1-year intervention period plus 3-year follow-

up period), with a range of 3-5 years. The Regenstrief programmer who worked on our IMPACT study<sup>35</sup> will identify candidate CVD events by searching the INPC every 6 months (blind to assignment), with the last search performed on the end date. To capture the small number of events that may occur outside of the INPC catchment area, patients will complete a CVD questionnaire at mid- and post-treatment and during the follow-up calls. If a reported event is not in the INPC, we will request medical records from the patient to confirm the event. Our cardiologist (Dr. Kovacs), also blinded, will use standardized criteria to adjudicate all CVD events for this exploratory outcome. Dr. Kovacs has served on endpoint committees for past trials. When needed, Dr. Kovacs will consult with the cardiologist on the DSMB (also blinded). Given that we are coding "harder" events and that many events will be positive for multiple markers, it is unlikely that coded events will be misclassified. We may fail to detect (and thus initially misclassify) a few events through INPC, which is why we are obtaining patient reports and medical records.

# Atherogenic Behavioral Factors

The BRFSS Tobacco Use Questionnaire, International Physical Activity Questionnaire, and the Morisky Questionnaire (MMAS-8) will assess tobacco use, physical activity, and adherence to cholesterol and blood pressure medications, respectively. Each scale possesses strong psychometric properties. 196-198

#### Conventional CVD Risk Factors

SBP and DBP will be the mean of the last 2 of 3 readings. Fasting cholesterol, glucose, insulin, and HbA1c will be quantified using standard methods. BMI will be computed from measured height and weight.

#### Miscellaneous Factors

Standard questions from our pilot studies will be used to assess demographics, medical history/update, psychiatric history/update, and current medications. Depression care variables (e.g., dose and duration of antidepressants, # and type of psychotherapy sessions) will be extracted from the treatment notes for eIMPACT patients. To obtain additional depression care data, all patients will complete a brief interview at the mid- and post-treatment visits and during the follow-up calls. Consistent with approved Authorization Form for this study, we will also periodically extract relevant depression treatment data (e.g., dose and duration of antidepressants) from the electronic medical record for all patients. We will also assess anxiety symptoms using the Generalized Anxiety Disorder-7 (GAD-7),<sup>200</sup> hostility/anger using the Buss-Perry Aggression Questionnaire,<sup>201</sup> trait positive affect using the Positive Affect subscale of the Positive and Negative Affect Schedule (PANAS),<sup>202,203</sup> and sleep quality using the Pittsburgh Sleep Quality Index,<sup>203</sup> all of which are widely used and validated instruments. We will also assess depression treatment satisfaction using an item employed in other recent depression trials conducted on the IUPUI campus and for the occurrence of any potential adverse events using a brief questionnaire. Finally, the Regenstrief programmer will identify potential adverse events by searching the INPC every 6 months (before DSMB meetings) for emergency department visits, hospitalizations, and deaths.

All items of the questionnaires to be administered at the pre-treatment visit (see Appendix 2), mid-treatment visit (see Appendix 3), post-treatment visit (see Appendix 4), and annual follow-up calls (see Appendix 5) can be found in the appendices.

#### Suicidal Ideation Protection Protocol

For the entire protocol, see Appendix 6.

### 6.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

We have developed a Data and Safety Monitoring Plan and Board to ensure the safety of participants and to monitor data quality and participant recruitment, accrual, and retention.

### Data and Safety Monitoring Plan:

- If an adverse event occurs, its severity will be promptly graded using the following scale:
  - 1. Mild: Awareness of sign or symptom but easily tolerated
  - 2. Moderate: Interference with normal daily activities
  - 3. Severe: Inability to perform normal daily activities

- 4. Life Threatening: Immediate risk of death from the reaction as it occurred
- After grading severity, the attribution of the adverse event will be graded using the following scale:
  - 1. Definite: Adverse event clearly related to study involvement
  - 2. Probable: Adverse event likely related to study involvement
  - 3. Possible: Adverse event may be related to study involvement
  - 4. Unlikely: Adverse event doubtfully related to study involvement
  - 5. Unrelated: Adverse event clearly not related to study involvement
- All adverse events that meet the IUPUI IRB prompt reporting requirements (i.e., unexpected, related or
  possibly related to participation in the research, and suggest that the research places subjects or others
  at a greater risk of harm than was previously known or recognized) will be reported the IUPUI IRB,
  CRC Research Subject Advocate, and NIH immediately. All other adverse events will be reported to
  these entities at the time of continuing review.
- A summary of adverse event data (frequency, types, and corrective actions) will be provided to the IUPUI IRB, CRC Research Subject Advocate, and NIH at the time of continuing review.

#### Data and Safety Monitoring Board:

- A 4-member, independent Data and Safety Monitoring Board (DSMB) will be formed to provide
  independent oversight. The DSMB will consist of a psychiatrist (from the Indiana University Department
  of Psychiatry), a cardiologist (from the Indiana University Krannert Institute of Cardiology), a clinical
  trialist (from the Indiana University Department of Biostatistics), and a medical ethicist (from the Indiana
  University Center for Aging Research), all of whom will not be part of the study team.
- Adverse events that are severe, life-threatening, or unanticipated will be immediately reviewed by the DSMB. At 6-month intervals, the DSMB will prepare a formal report of participant recruitment, accrual, retention, data quality, and adverse events. At that time, the DSMB will also determine whether the study should continue unchanged, be modified, or be stopped. The IUPUI IRB, CRC Research Subject Advocate, and NIH will receive copies of all DSMB reports at the time of continuing review.

# 7.0 Study Withdrawal/Discontinuation

All participants will be considered enrolled at the end of the ResNet interview. The informed consent statement describes the possibility of and the procedures for withdrawing from the study. A participant may notify either the principal investigator or any member of the research team at any time via email, phone, or in-person that s/he wants to withdraw from the study for any reason. The schedule of participant reimbursement is as follows: \$100 for the pre-treatment visit, \$25 for the mid-treatment call, \$100 for the post-treatment visit, \$20 for each of the annual follow-up calls, and up to \$10 per visit to cover parking or transportation costs. If a participant withdraws before the pre-treatment assessment visit, no payment will be provided.

Other reasons for study withdrawal/discontinuation are (a) the participant's primary care provider or another provider seeing the participant (e.g., a psychiatrist outside of the study team) no longer believes that his/her patient is appropriate for this trial after a triggering of the Suicidal Ideation Protection Protocol or any other reason, (b) the participant develops acute or serious illness that precludes completion of the main study visits within the allowed timeframes, and (c) the participant, in the assessment of the eIMPACT psychiatrist, exhibits evidence of a psychotic disorder or bipolar disorder (both of which are exclusionary conditions and could interfere with treatment delivery/effectiveness) during the 1-year treatment phase of the trial. In the case of situation (b), the patient will not complete any future study visits or calls. However, if the patient provides permission, electronic medical record data (e.g., incident CVD events) will still be obtained going forward, consistent with our Authorization Form. In the case of situation (c), patients with a psychotic disorder or bipolar disorder would likely benefit from psychotropic medications, such as antipsychotic medications or mood stabilizer, that are beyond what are provided in this trial.

For Usual Care patients who score in the "severe depression" range (20-27) on the PHQ-9 at the midtreatment (6 months), the DCS (a) will contact the patient's primary care provider in person, by phone, or through the electronic medical record to notify the provider of the patient's high depressive symptoms and to urge the provider to follow-up and (b) will provide a list of local mental health services, including referral to a psychiatrist outside of the study team. In addition, participants in both treatment groups who continue to exhibit

elevated depressive symptoms (PHQ-9 ≥10) at post-treatment will be will urged to follow-up with their primary care providers regarding their depression. Their providers will also receive a letter from the study team indicating that their patient has completed participation in the treatment phase of the trial and continues to have elevated depressive symptoms. This letter will also urge physicians to follow-up with their patients and will provide a list of local mental health services. Finally, for participants in both treatment groups who score in the "severe depression" range (20-27) on the PHQ-9 during an annual follow-up call, the DCS (a) will contact the patient's primary care provider in person, by phone, or through the electronic medical record to notify the provider of the patient's high depressive symptoms and to urge the provider to follow-up and (b) will provide a list of local mental health services, including referral to a psychiatrist outside of the study team.

#### 8.0 Statistical Considerations

# Sample Size and Power Considerations

# Endothelial Dysfunction

Using the effect size of depression treatment on FMD from our pilot trial, we need 88 patients (44 per arm) to detect a group difference in FMD of 1.7% (d = 0.61) at 12 months, assuming a power level of 0.80 and a Type I error of 0.05. This would be a clinically relevant difference. Assuming a conservative attrition rate of 20%, <sup>204</sup> we will have 172 completers (220 x .80) for FMD, yielding power levels of 0.98 for d = 0.61 and 0.80 for d = 0.43.

#### Candidate Mechanisms

We expect at a power level  $\geq$ 0.80 for the candidate mechanisms (Hypotheses 2-5), as we will be able to detect effect sizes as small as d = 0.43 with 172 completers. In our IMPACT study<sup>35</sup> and pilot trial, effect sizes for depressive symptoms (d = 0.69 and 1.33), IL-6 (d = 0.43), and CRP (d = 0.78) were in the medium-to-large range. In other studies, effect sizes of 0.52 were found for psychological interventions on heart rate variability, <sup>205-207</sup> 1.00 for SSRIs on IL-6, <sup>143</sup> 0.74 for SSRIs <sup>143</sup> and 0.85 for CBT<sup>138</sup> on CRP, 0.91<sup>146</sup> and 0.46<sup>144</sup> for SSRIs on BTG, and 0.87 for SSRIs on PF4. <sup>144</sup>

# CVD Events

Over the mean observation period of 4 years, we anticipate a cumulative CVD event rate of 20% (39 events) and a 25% lower relative risk (HR ≤ 0.75) in elMPACT versus usual care. These estimates are reasonable, as we observed a CVD event rate of 24% and a 46% lower relative risk (event rate: 18% vs. 31%) in our IMPACT secondary analysis that had a 4-year observation period. Our high-risk sample will differ from the typical sample of a risk reduction trial in that (a) all patients will have depression and ≥1 CVD risk factor and (b) many will be of low SES and/or African American, two groups at elevated risk for CVD event.<sup>1,171</sup> Although we expect to have CVD event data for nearly all patients, we assume a conservative attrition rate of 10%, leaving 194 completers. As is typical of Phase 2 trials, our trial is not designed to detect a statistically significant difference in clinical events; however, a 25% relative risk reduction would be a clinically relevant signal (statin therapy reduces risk by ≈30%<sup>156</sup>) and has been used to power recent event-driven Phase 3 cardiology trials.<sup>157</sup>

#### Statistical Analyses

We will use the intent-to-treat approach.  $^{208}$  All tests will be two-tailed with p < .05 considered significant. Supplemental analyses of completers will be performed. We will assess for differences in all baseline factors. Due to randomization, we do not expect baseline group differences. Even so, any differences will be taken into account when interpreting results, and any baseline factors that differ between the groups will be included as covariates in sensitivity analyses. Aim 1: We will test our hypothesis that eIMPACT patients will exhibit greater improvement in endothelial dysfunction (Hypothesis 1) by performing a two-sample t-test with FMD at 12 months as the dependent variable. If there is a group difference in baseline FMD, analyses of covariance (ANCOVAs) adjusting for baseline level will also be performed. We will also explore whether eIMPACT patients show a clinically relevant reduction (25% lower relative risk) in CVD events by running a Cox proportional hazards model with treatment group predicting time to first CVD event. Patients will be censored at non-CVD death or the end date. We expect to observe a HR  $\leq$  0.75. Aim 2. We will test our hypotheses that eIMPACT patients will exhibit greater decreases in the candidate mechanisms (Hypotheses 2-5) by performing two-sample t-tests with SCL-20 score, high-frequency heart rate variability, IL-6, CRP, BTG, and PF4 at 12 months as the dependent variables. If baseline group differences are found, ANCOVAs adjusting for baseline level will Revision Date: July 13, 2018

also be performed. To explore whether decreases in the candidate mechanisms are associated with improvements in endothelial dysfunction, we will compute correlations between 12-month change in each mechanism and in FMD. To explore whether decreases in the candidate mechanisms are partial mediators of eIMPACT's hypothesized cardioprotective effect, we will conduct exploratory mediation analyses using MacKinnon's approach, which has greater power than others.<sup>209</sup> First, to quantify the treatment effect on each mechanism ("a" coefficients), we will perform linear regressions with treatment group predicting 12-month level of each mechanism. Second, to quantify the effect of each candidate mechanism on endothelial dysfunction ("b" coefficients), we will perform linear regressions with 12-month level of each mechanism predicting 12-month FMD in the presence of treatment group. Third, the significance of each mediation effect will be tested using MacKinnon and Lockwood's product of coefficients ("ab") method employing asymmetric confidence limits.<sup>209,210</sup> If this test is significant, the selected mechanism is a partial mediator of the treatment effect on 12-month FMD. Of note, we will also explore (a) if changes in depressive symptoms are correlated with changes in the atherogenic physiologic factors and (b) if changes in FMD predict CVD events.

# Supplemental, Hypothesis-Generating Analyses

(1) We will explore atherogenic behavioral factors, conventional CVD risk factors, and depression care variables as potential mechanisms of elMPACT's effect on FMD by repeating Aim 2 analyses. (2) To explore the separate effects of intervention components (which likely have shared and unique pathways; Figure 1), Aim 1 and 2 analyses will be repeated after coding the treatment variable as follows: elMPACT both components, elMPACT antidepressants only, elMPACT psychotherapy only, elMPACT neither component, and usual care. (3) We will explore sex and race/ethnicity as moderators of the treatment effect on the outcomes. (4) We will estimate the cost per patient of providing elMPACT, including charges for BtB, DCS, psychiatrist and primary care expert supervision, materials, and a telephone line.

# 9.0 Privacy/Confidentiality Issues

Participants will be screened and consented in the privacy of their homes via telephone and/or in private rooms at the targeted primary care clinics or the CRC. All procedures will take place in private rooms at the CRC, Dr. Stewart's Cardiovascular Behavioral Medicine Laboratory, the targeted primary care clinics, or a location selected by the patient, such as their home or a family member's/friend's home (for the follow-up calls and the telephonic and computerized components of the elMPACT intervention). All research material will be kept strictly confidential. All study personnel have completed Collaborative Institutional Training Initiative (CITI) courses in human subjects research and will make every effort to ensure confidentiality. All electronic and hard copy data will be identified using only the unique participant number assigned when each individual is enrolled in this study (participant identifying information will not be included). All electronic data will be saved on password-protected and encrypted computers and secure servers, and all hard copy data will be stored in secure and locked file cabinets. The key linking participant names with the participant numbers will be kept in a separate secure and locked file cabinet. Data will be analyzed and reported as an aggregate, with no individual identifying information.

# 10.0 Follow-Up and Record Retention

For Usual Care patients who score in the "severe depression" range (20-27) on the PHQ-9 at the midtreatment (6 months) or post-treatment (12 months) assessments, the DCS (a) will contact the patient's primary care provider in person or by phone to notify the provider of the patient's high depressive symptoms and to urge the provider to follow-up and (b) will provide a list of local mental health services, including referral to a psychiatrist outside of the study team. In addition, participants in both treatment groups who continue to exhibit elevated depressive symptoms (PHQ-9 ≥10) at post-treatment will be will urged to follow-up with their primary care providers regarding their depression. Their providers will also receive a letter from the study team indicating that their patient has completed participation in the treatment phase of the trial and continues to have elevated depressive symptoms. This letter will also urge physicians to follow-up with their patients and will provide a list of local mental health services.

While the study duration is five years, all study documents will be kept up to seven years after study completion. After this time, we will permanently delete patient identifying data and shred all paper records, per Indiana State law. This process prevents any opportunity for a breach of confidentiality to occur.

#### **Literature Cited**

- 1. Go AS, Mozaffarian D, Roger VL, et al. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. *Circulation*. 2013;127(1):e6-e245.
- 2. Hoyert D, Xu J. Deaths: preliminary data for 2011. *National Vital Statistics Reports*. 2012;61(6).
- 3. Kessler RC, Berglund P, Demler O, et al. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). *JAMA*. Jun 18 2003;289(23):3095-3105.
- 4. Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. *JAMA*. Nov 10 1999;282(18):1737-1744.
- 5. Spitzer RL, Williams JB, Kroenke K, et al. Utility of a new procedure for diagnosing mental disorders in primary care. The PRIME-MD 1000 study. *JAMA*. Dec 14 1994;272(22):1749-1756.
- 6. Murray CJ, Lopez AD. The global burden of disease: A comprehensive assessment of mortality and disability from disease, injuries and risk factors in 1990 and projected to 2020 Boston, MA: Harvard School of Public Health on behalf of the World Health Organization and the World Bank; 1996.
- 7. Greenberg PE, Kessler RC, Birnbaum HG, et al. The economic burden of depression in the United States: how did it change between 1990 and 2000? *J Clin Psychiatry*. Dec 2003;64(12):1465-1475.
- 8. Van der Kooy K, van Hout H, Marwijk H, Marten H, Stehouwer C, Beekman A. Depression and the risk for cardiovascular diseases: systematic review and meta analysis. *International Journal of Geriatric Psychiatry*. Jul 2007;22(7):613-626.
- 9. Meijer A, Conradi HJ, Bos EH, Thombs BD, van Melle JP, de Jonge P. Prognostic association of depression following myocardial infarction with mortality and cardiovascular events: a meta-analysis of 25 years of research. *General Hospital Psychiatry*. May-Jun 2011;33(3):203-216.
- 10. Rugulies R. Depression as a predictor for coronary heart disease. a review and meta-analysis. *American Journal of Preventive Medicine*. 2002;23(1):51-61.
- 11. Wulsin LR, Singal BM. Do depressive symptoms increase the risk for the onset of coronary disease? A systematic quantitative review. *Psychosom Med.* Mar-Apr 2003;65(2):201-210.
- 12. Rozanski A, Blumenthal JA, Davidson KW, Saab PG, Kubzansky L. The epidemiology, pathophysiology, and management of psychosocial risk factors in cardiac practice: the emerging field of behavioral cardiology. *Journal of the American College of Cardiology*. 2005;45(5):637-651.
- 13. Brown JM, Stewart JC, Stump TE, Callahan CM. Risk of coronary heart disease events over 15 years among older adults with depressive symptoms. *Am J Geriatr Psychiatry*. Aug 2011;19(8):721-729.
- 14. Rosengren A, Hawken S, Ôunpuu S, et al. Association of psychosocial risk factors with risk of acute myocardial infarction in 11 119 cases and 13 648 controls from 52 countries (the INTERHEART study): Case-control study. *Lancet*. 2004;364:953-962.
- 15. Stewart JC, Zielke DJ, Hawkins MA, et al. Depressive symptom clusters and 5-year incidence of coronary artery calcification: the coronary artery risk development in young adults study. *Circulation*. Jul 24 2012;126(4):410-417.
- 16. Suls J, Bunde J. Anger, anxiety, and depression as risk factors for cardiovascular disease: the problems and implications of overlapping affective dispositions. *Psychological Bulletin*. 2005;131(2):260-300.
- 17. Stewart JC, Janicki DL, Muldoon MF, Sutton-Tyrrell K, Kamarck TW. Negative emotions and 3-year progression of subclinical atherosclerosis. *Arch Gen Psychiatry*. 2007;64(2):225-233.
- 18. Hill AB. The environment and disease: Association or causation? *Proceedings of the Royal Society of Medicine*. 1965;58:295-300.
- 19. Shively CA, Register TC, Adams MR, Golden DL, Willard SL, Clarkson TB. Depressive behavior and coronary artery atherogenesis in adult female cynomolgus monkeys. *Psychosom Med.* Jul 2008;70(6):637-645.
- 20. McCaffery JM, Frasure-Smith N, Dube MP, et al. Common genetic vulnerability to depressive symptoms and coronary artery disease: a review and development of candidate genes related to inflammation and serotonin.[see comment]. *Psychosom Med.* 2006;68(2):187-200.
- 21. Berkman LF, Blumenthal J, Burg M, et al. Effects of treating depression and low perceived social support on clinical events after myocardial infarction: the Enhancing Recovery in Coronary Heart Disease Patients (ENRICHD) Randomized Trial. *JAMA*. 2003;289(23):3106-3116.
- 22. Glassman AH, O'Connor CM, Califf RM, et al. Sertraline treatment of major depression in patients with acute MI or unstable angina. *JAMA*. 2002;288(6):701-709.

- 23. van Melle JP, de Jonge P, Honig A, et al. Effects of antidepressant treatment following myocardial infarction. *British Journal of Psychiatry*. 2007;190:460-466.
- 24. Carney RM, Freedland KE. Treatment-resistant depression and mortality after acute coronary syndrome. *Am J Psychiatry*. Apr 2009;166(4):410-417.
- 25. Glassman AH, Bigger JT, Jr., Gaffney M. Psychiatric characteristics associated with long-term mortality among 361 patients having an acute coronary syndrome and major depression: seven-year follow-up of SADHART participants. *Arch Gen Psychiatry*. Sep 2009;66(9):1022-1029.
- 26. Zuidersmaa M, Conradia HJ, van Melle JP, Ormela J, de Jonge P. Depression treatment after myocardial infarction and long-term risk of subsequent cardiovascular events and mortality: A randomized controlled trial. *J Psychosom Res.* 2013;74(1):25-30.
- 27. de Jonge P, Honig A, van Melle JP, et al. Nonresponse to treatment for depression following myocardial infarction: association with subsequent cardiac events. *Am J Psychiatry*. Sep 2007;164(9):1371-1378.
- 28. Shapiro PA. Depression treatment and coronary artery disease outcomes: Time for reflection. *J Psychosom Res.* 2013;74(1):4-5.
- 29. Ziegelstein RC. Improving depression and reducing cardiac events: Which is the chicken and which is the egg? *J Psychosom Res.* 2013;74(5):454-457.
- 30. Katon WJ, Lin EH, Von Korff M, et al. Collaborative care for patients with depression and chronic illnesses. *N Engl J Med.* Dec 30 2010;363(27):2611-2620.
- 31. Davidson KW, Rieckmann N, Clemow L, et al. Enhanced depression care for patients with acute coronary syndrome and persistent depressive symptoms: coronary psychosocial evaluation studies randomized controlled trial. *Archives of Internal Medicine*. 2010;170(7):600-608.
- 32. Ye S, Shaffer JA, Rieckmann N, et al. Long-term outcomes of enhanced depression treatment in patients with acute coronary syndromes. *Am J Med.* May 14 2014.
- 33. Shimbo D, Davidson KW, Haas DC, Fuster V, Badimon JJ. Negative impact of depression on outcomes in patients with coronary artery disease: mechanisms, treatment considerations, and future directions. *Journal of Thrombosis & Haemostasis*. 2005;3(5):897-908.
- 34. Goldston K, Baillie AJ. Depression and coronary heart disease: A review of epidemiological evidence, explanatory mechanisms, and management approaches. *Clinical Psychology Review*. 2008;28:288-306.
- 35. Stewart JC, Perkins AJ, Callahan CM. Effect of collaborative care for depression on risk of cardiovascular events: data from the IMPACT randomized controlled trial. *Psychosom Med.* 2014;76:29-37.
- 36. Unutzer J, Katon W, Callahan CM, et al. Collaborative care management of late-life depression in the primary care setting: a randomized controlled trial. *JAMA*. 2002;288(22):2836-2845.
- 37. Ali S, Stone MA, Peters JL, Davies MJ, Khunti K. The prevalence of co-morbid depression in adults with Type 2 diabetes: a systematic review and meta-analysis. *Diabet Med.* Nov 2006;23(11):1165-1173.
- 38. Rabkin JG. HIV and depression: 2008 review and update. Curr HIV/AIDS Rep. Nov 2008;5(4):163-171.
- 39. National Heart L, and Blood Institute. Shaping the future of research: a strategic plan for the National Heart, Lung, and Blood Institute.

  <a href="http://www.nhlbi.nih.gov/about/strategicplan/documents/StrategicPlan Appendix.pdf">http://www.nhlbi.nih.gov/about/strategicplan/documents/StrategicPlan Appendix.pdf</a>. Accessed May 20, 2013.
- 40. Lorant V, Deliege D, Eaton W, Robert A, Philippot P, Ansseau M. Socioeconomic inequalities in depression: a meta-analysis. *Am J Epidemiol*. Jan 15 2003;157(2):98-112.
- 41. Ference BA, Yoo W, Alesh I, et al. Effect of long-term exposure to lower low-density lipoprotein cholesterol beginning early in life on the risk of coronary heart disease: a Mendelian randomization analysis. *Journal of the American College of Cardiology*. Dec 25 2012;60(25):2631-2639.
- 42. Law MR, Wald NJ, Rudnicka AR. Quantifying effect of statins on low density lipoprotein cholesterol, ischaemic heart disease, and stroke: systematic review and meta-analysis. *BMJ*. 2003;326(7404):1423.
- 43. Law MR, Wald NJ, Thompson SG. By how much and how quickly does reduction in serum cholesterol concentration lower risk of ischaemic heart disease? *BMJ*. Feb 5 1994;308(6925):367-372.
- 44. Rodenburg J, Vissers MN, Wiegman A, et al. Statin treatment in children with familial hypercholesterolemia: the younger, the better. *Circulation*. Aug 7 2007;116(6):664-668.
- 45. Domanski M, Lloyd-Jones D, Fuster V, Grundy S. Can we dramatically reduce the incidence of coronary heart disease? *Nat Rev Cardiol.* 2011;8(12):721-725.

- 46. Domanski MJ. Primary prevention of coronary artery disease. *N Engl J Med.* Oct 11 2007;357(15):1543-1545.
- 47. McGill HC, Jr., McMahan CA. Starting earlier to prevent heart disease. *JAMA*. Nov 5 2003;290(17):2320-2322.
- 48. Steinberg D. Earlier intervention in the management of hypercholesterolemia: what are we waiting for? *Journal of the American College of Cardiology.* Aug 17 2010;56(8):627-629.
- 49. Steinberg D, Glass CK, Witztum JL. Evidence mandating earlier and more aggressive treatment of hypercholesterolemia. *Circulation*. Aug 5 2008;118(6):672-677.
- 50. Steinberg D, Grundy SM. The case for treating hypercholesterolemia at an earlier age: moving toward consensus. *Journal of the American College of Cardiology*. Dec 25 2012;60(25):2640-2642.
- 51. Cooper DC, Tomfohr LM, Milic MS, et al. Depressed mood and flow-mediated dilation: a systematic review and meta-analysis. *Psychosom Med.* Jun 2011;73(5):360-369.
- 52. Ell K, Xie B, Quon B, Quinn DI, Dwight-Johnson M, Lee PJ. Randomized controlled trial of collaborative care management of depression among low-income patients with cancer. *Journal of Clinical Oncology*. 2008;26(27):4488-4496.
- 53. Janssen I, Powell LH, Matthews KA, et al. Depressive symptoms are related to progression of coronary calcium in midlife women. *American Heart Journal*. 2011;161(6):1186-1191.
- 54. Thombs BD, de Jonge P, Coyne JC, et al. Depression screening and patient outcomes in cardiovascular care: a systematic review. *JAMA*. 2008;300(18):2161-2171.
- 55. Alexopoulos GS, Meyers BS, Young RC, Campbell S, Silbersweig D, Charlson M. The "vascular depression" hypothesis. *Arch Gen Psychiatry*. Oct 1997;54(10):915-922.
- O'Brien J, Ames D, Chiu E, Schweitzer I, Desmond P, Tress B. Severe deep white matter lesions and outcome in elderly patients with major depressive disorder: follow up study. *Br Med J*. 1998;317(7164):982-984.
- 57. Simpson S, Baldwin RC, Jackson A, Burns AS. Is subcortical disease associated with a poor response to antidepressants? Neurological, neuropsychological and neuroradiological findings in late-life depression. *Psychological Medicine*. 1998;28(5):1015-1026.
- 58. Lesperance F, Frasure-Smith N, Talajic M. Major depression before and after myocardial infarction: its nature and consequences. *Psychosom Med.* 1996;58(2):99-110.
- 59. Schleifer SJ, Macari-Hinson MM, Coyle DA, et al. The nature and course of depression following myocardial infarction. *Archives of Internal Medicine*. 1989;149(8):1785-1789.
- 60. Davidson KW, Bigger JT, Burg MM, et al. Centralized, stepped, patient preference-based treatment for patients with post-acute coronary syndrome depression: CODIACS Vanguard randomized controlled trial. *JAMA Intern Med.* Mar 7 2013:1-8.
- 61. Scheier MF, Bridges MW. Person variables and health: personality predispositions and acute psychological states as shared determinants for disease. *Psychosom Med.* May-Jun 1995;57(3):255-268.
- 62. Elderon L, Whooley MA. Depression and Cardiovascular Disease. *Progress in Cardiovascular Diseases*. 2013;55(6):511-523.
- 63. Rollman BL, Belnap BH, LeMenager MS, et al. Telephone-delivered collaborative care for treating post-CABG depression: A randomized controlled trial. *JAMA*. 2009;302(19):2095-2103.
- 64. Unutzer J, Katon W, Williams JW, Jr., et al. Improving primary care for depression in late life: the design of a multicenter randomized trial. *Medical Care*. 2001;39(8):785-799.
- 65. Unutzer J, investigators tl. *IMPACT Intervention Manual*. Los Angeles, CA: Center for Health Services Research, UCLA Neuropsychiatric Institute;1999.
- 66. Marks IM, Cavanagh K, Gega L. *Hands-on Help: Computer-aided Psychotherapy.* Hove, UK: Psychology Press; 2007.
- 67. Proudfoot J, Goldberg D, Mann A, Everitt B, Marks I, Gray JA. Computerized, interactive, multimedia cognitive-behavioural program for anxiety and depression in general practice. *Psychological Medicine*. 2003;33(2):217-227.
- 68. Proudfoot J, Ryden C, Everitt B, et al. Clinical efficacy of computerised cognitive-behavioural therapy for anxiety and depression in primary care: randomised controlled trial. *British Journal of Psychiatry*. 2004;185:46-54.
- 69. Grime P. Computerized cognitive behavioural therapy at work: A randomized controlled trial in employees with recent stress-related absenteeism. *Occupational Medicine*. 2003;53:538.

- 70. Hunt S, Howells E, Stapleton B. The addition of computerised CBT program to a stepped care, primary care mental health service. *Journal of Primary Care Mental Health*. 2006;9:34-38.
- 71. Learmonth D, Learmonth D, Trosh J, Rai S, Sewell J, Cavanagh K. The role of computer-aided psychotherapy within an NHS CBT specialist service. *Counselling & Psychotherapy Research*. 2008;8(2):117.
- 72. Learmonth D, Rai S. Establishing the effectiveness of computerised cognitive behavioral therapy for secondary/tertiary mental health care service users with and without physical co-morbidities. *Health Psychology Update*. 2007;16:42-48.
- 73. Learmonth D, Rai S. Taking computerized CBT beyond primary care. *British Journal of Clinical Psychology*. 2008;47(Pt 1):111-118.
- 74. Mitchell N, Dunn K. Pragmatic evaluation of the viability of CCBT self-help for depression in higher education. *Counseling & Psychotherapy Research*. 2007;7:144-150.
- van den Berg S, Shapiro DA, Bickerstaffe D, Cavanagh K. Computerized cognitive-behaviour therapy for anxiety and depression: a practical solution to the shortage of trained therapists. *Journal of Psychiatric & Mental Health Nursing*. 2004;11(5):508-513.
- 76. Gloaguen V, Cottraux J, Cucherat M, Blackburn IM. A meta-analysis of the effects of cognitive therapy in depressed patients. *Journal of Affective Disorders*. 1998;49:59-72.
- 77. McMurchie W, Macleod F, Power K, Laidlaw K, Prentice N. Computerised cognitive behavioural therapy for depression and anxiety with older people: a pilot study to examine patient acceptability and treatment outcome. *International Journal of Geriatric Psychiatry*. Nov 2013;28(11):1147-1156.
- 78. NICE. Computerised cognitive behavioural therapy (CCBT) for the treatment of depression and anxiety. Technology Appraisal no. 97. London: NICE;2006.
- 79. McHugh R, Santucci L, Elkins R, Schechter B, Barlow DH. Effectiveness of computerized CBT in a university health setting. 2010 World Congress of Behavioral and Cognitive Therapies; June, 2010.
- 80. NICE. Computerised cognitive behavioural therapy (CCBT) for the treatment of depression and anxiety: Costing report and costing template. Technology Appraisal no. 97. London: NICE;2006.
- 81. Corretti MC, Anderson TJ, Benjamin EJ, et al. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. *Journal of the American College of Cardiology*. 2002;39(2):257-265.
- 82. Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999;340(2):115-126.
- 83. Celermajer DS, Sorensen KE, Gooch VM, et al. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. *Lancet*. 1992;340(8828):1111-1115.
- 84. Takase B, Uehata A, Akima T, et al. Endothelium-dependent flow-mediated vasodilation in coronary and brachial arteries in suspected coronary artery disease. *Am J Cardiol.* Dec 15 1998;82(12):1535-1539. A1537-1538.
- 85. Anderson TJ, Uehata A, Gerhard MD, et al. Close relation of endothelial function in the human coronary and peripheral circulations. *J. Am. Coll. Cardiol.* Nov 1 1995;26(5):1235-1241.
- 86. Vogel RA. Measurement of endothelial function by brachial artery flow-mediated vasodilation. *Am J Cardiol.* Jul 19 2001;88(2A):31E-34E.
- 87. Flammer AJ, Anderson T, Celermajer DS, et al. The assessment of endothelial function: from research into clinical practice. *Circulation*. Aug 7 2012;126(6):753-767.
- 88. Frick M, Weidinger F. Endothelial function: a surrogate endpoint in cardiovascular studies? *Curr Pharm Des.* 2007:13(17):1741-1750.
- 89. Vita JA, Keaney JF, Jr. Endothelial function: a barometer for cardiovascular risk? *Circulation*. Aug 6 2002;106(6):640-642.
- 90. Antony I, Aptecar E, Lerebours G, Nitenberg A. Coronary artery constriction caused by the cold pressor test in human hypertension. *Hypertension*. 1994;24(2):212-219.
- 91. Benjamin EJ, Larson MG, Keyes MJ, et al. Clinical correlates and heritability of flow-mediated dilation in the community: the Framingham Heart Study. *Circulation*. 2004;109(5):613-619.
- 92. Celermajer DS, Sorensen KE, Bull C, Robinson J, Deanfield JE. Endothelium-dependent dilation in the systemic arteries of asymptomatic subjects relates to coronary risk factors and their interaction. *Journal of the American College of Cardiology*. 1994;24(6):1468-1474.
- 93. Rubenfire M, Rajagopalan S, Mosca L. Carotid artery vasoreactivity in response to sympathetic stress correlates with coronary disease risk and is independent of wall thickness. *Journal of the American College of Cardiology.* 2000;36(7):2192-2197.

- 94. Treasure CB, Manoukian SV, Klein JL, et al. Epicardial coronary artery responses to acetylcholine are impaired in hypertensive patients. *Circulation Research*. 1992;71(4):776-781.
- 95. Vita JA, Treasure CB, Nabel EG, et al. Coronary vasomotor response to acetylcholine relates to risk factors for coronary artery disease. *Circulation*. 1990;81(2):491-497.
- 96. Zeiher AM, Drexler H, Wollschlager H, Just H. Modulation of coronary vasomotor tone in humans. Progressive endothelial dysfunction with different early stages of coronary atherosclerosis. *Circulation*. 1991;83(2):391-401.
- 97. Witte DR, Westerink J, de Koning EJ, van der Graaf Y, Grobbee DE, Bots ML. Is the association between flow-mediated dilation and cardiovascular risk limited to low-risk populations? *Journal of the American College of Cardiology*. 2005;45(12):1987-1993.
- 98. Enderle MD, Schroeder S, Ossen R, et al. Comparison of peripheral endothelial dysfunction and intimal media thickness in patients with suspected coronary artery disease. *Heart.* 1998;80(4):349-354.
- 99. Neunteufl T, Katzenschlager R, Hassan A, et al. Systemic endothelial dysfunction is related to the extent and severity of coronary artery disease. *Atherosclerosis*. 1997;129(1):111-118.
- 100. Juonala M, Viikari JS, Laitinen T, et al. Interrelations between brachial endothelial function and carotid intima-media thickness in young adults: the cardiovascular risk in young Finns study. *Circulation*. 2004;110(18):2918-2923.
- 101. Fichtlscherer S, Breuer S, Zeiher AM. Prognostic value of systemic endothelial dysfunction in patients with acute coronary syndromes: further evidence for the existence of the "vulnerable" patient. *Circulation*. 2004;110(14):1926-1932.
- 102. Gokce N, Keaney JF, Jr., Hunter LM, et al. Predictive value of noninvasively determined endothelial dysfunction for long-term cardiovascular events in patients with peripheral vascular disease. *Journal of the American College of Cardiology*. 2003;41(10):1769-1775.
- 103. Halcox JP, Schenke WH, Zalos G, et al. Prognostic value of coronary vascular endothelial dysfunction. *Circulation*. 2002;106(6):653-658.
- 104. Heitzer T, Schlinzig T, Krohn K, Meinertz T, Munzel T. Endothelial dysfunction, oxidative stress, and risk of cardiovascular events in patients with coronary artery disease. *Circulation*. 2001;104(22):2673-2678.
- 105. Neunteufl T, Heher S, Katzenschlager R, et al. Late prognostic value of flow-mediated dilation in the brachial artery of patients with chest pain. *Am J Cardiol*. 2000;86(2):207-210.
- 106. Perticone F, Ceravolo R, Pujia A, et al. Prognostic significance of endothelial dysfunction in hypertensive patients. *Circulation*. 2001;104(2):191-196.
- 107. Rossi R, Nuzzo A, Origliani G, et al. Prognostic role of flow-mediated dilation and cardiac risk factors in post-menopausal women. *Journal of the American College of Cardiology*. Mar 11 2008;51(10):997-1002.
- 108. Schachinger V, Britten MB, Zeiher AM. Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease. *Circulation*. 2000;101(16):1899-1906.
- 109. Schindler TH, Hornig B, Buser PT, et al. Prognostic value of abnormal vasoreactivity of epicardial coronary arteries to sympathetic stimulation in patients with normal coronary angiograms. *Arteriosclerosis, Thrombosis & Vascular Biology.* 2003;23(3):495-501.
- 110. Shimbo D, Grahame-Clarke C, Miyake Y, et al. The association between endothelial dysfunction and cardiovascular outcomes in a population-based multi-ethnic cohort. *Atherosclerosis*. 2007;192(1):197-203.
- 111. Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR, Jr., Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. *Circulation*. 2000;101(9):948-954.
- 112. Yeboah J, Folsom AR, Burke GL, et al. Predictive value of brachial flow-mediated dilation for incident cardiovascular events in a population-based study: the multi-ethnic study of atherosclerosis. *Circulation*. 2009;120(6):502-509.
- 113. Modena MG, Bonetti L, Coppi F, Bursi F, Rossi R. Prognostic role of reversible endothelial dysfunction in hypertensive postmenopausal women. *Journal of the American College of Cardiology*. 2002;40(3):505-510.
- 114. Suessenbacher A, Frick M, Alber HF, Barbieri V, Pachinger O, Weidinger F. Association of improvement of brachial artery flow-mediated vasodilation with cardiovascular events. *Vascular Medicine*. 2006;11(4):239-244.

- 115. Kitta Y, Obata JE, Nakamura T, et al. Persistent impairment of endothelial vasomotor function has a negative impact on outcome in patients with coronary artery disease. *Journal of the American College of Cardiology.* Jan 27 2009;53(4):323-330.
- 116. Blaha MJ, Michos ED. Niacin--a case study for the role of event-driven versus surrogate endpoint trials. *Heart.* Nov 2013;99(22):1631-1632.
- 117. McDonald CJ, Overhage JM, Barnes M, et al. The Indiana network for patient care: a working local health information infrastructure. An example of a working infrastructure collaboration that links data from five health systems and hundreds of millions of entries. *Health Aff (Millwood)*. Sep-Oct 2005;24(5):1214-1220.
- 118. Biondich PG, Grannis SJ. The Indiana network for patient care: an integrated clinical information system informed by over thirty years of experience. *J Public Health Manag Pract.* Nov 2004;Suppl:S81-86
- 119. McDonald CJ, Overhage JM, Tierney WM, et al. The Regenstrief Medical Record System: a quarter century experience. *Int J Med Inform.* Jun 1999;54(3):225-253.
- 120. Carney RM, Freedland KE, Veith RC. Depression, the Autonomic Nervous System, and Coronary Heart Disease. *Psychosom Med.* May-Jun 2005;67(Suppl1):S29-S33.
- 121. DiMatteo MR, Lepper HS, Croghan TW. Depression Is a Risk Factor for Noncompliance With Medical Treatment Meta-analysis of the Effects of Anxiety and Depression on Patient Adherence. *Archives of Internal Medicine*. 2000;160(14):2101-2107.
- 122. Freedland KE, Carney RM, Skala JA. Depression and smoking in coronary heart disease. *Psychosom Med.* May-Jun 2005;67 Suppl 1:S42-46.
- 123. Joynt KE, Whellan DJ, O'Connor CM. Depression and cardiovascular disease: mechanisms of interaction. *Biological psychiatry*. Aug 1 2003;54(3):248-261.
- 124. Kop WJ, Gottdiener JS. The role of immune system parameters in the relationship between depression and coronary artery disease. *Psychosom Med.* May-Jun 2005;67(Suppl1):S37-S41.
- 125. Nemeroff CB, Musselman DL. Are platelets the link between depression and ischemic heart disease? *American Heart Journal.* Oct 2000;140(4 Suppl):57-62.
- 126. Patten SB, Williams JV, Lavorato DH, Eliasziw M. A longitudinal community study of major depression and physical activity. *General Hospital Psychiatry*. Nov-Dec 2009;31(6):571-575.
- 127. Carney RM, Blumenthal JA, Freedland KE, et al. Low heart rate variability and the effect of depression on post-myocardial infarction mortality. *Archives of Internal Medicine*. Jul 11 2005;165(13):1486-1491.
- 128. Kop WJ, Stein PK, Tracy RP, Barzilay JI, Schulz R, Gottdiener JS. Autonomic nervous system dysfunction and inflammation contribute to the increased cardiovascular mortality risk associated with depression. *Psychosom Med.* Sep 2010;72(7):626-635.
- 129. Surtees PG, Wainwright NW, Boekholdt SM, Luben RN, Wareham NJ, Khaw KT. Major depression, C-reactive protein, and incident ischemic heart disease in healthy men and women. *Psychosom Med.* Oct 2008;70(8):850-855.
- 130. Whooley MA, de Jonge P, Vittinghoff E, et al. Depressive symptoms, health behaviors, and risk of cardiovascular events in patients with coronary heart disease. *JAMA*. 2008;300(20):2379-2388.
- 131. Brummett BH, Babyak MA, Siegler IC, Mark DB, Williams RB, Barefoot JC. Effect of smoking and sedentary behavior on the association between depressive symptoms and mortality from coronary heart disease. *Am J Cardiol.* Sep 1 2003;92(5):529-532.
- 132. Win S, Parakh K, Eze-Nliam CM, Gottdiener JS, Kop WJ, Ziegelstein RC. Depressive symptoms, physical inactivity and risk of cardiovascular mortality in older adults: the Cardiovascular Health Study. *Heart.* Mar 2011;97(6):500-505.
- 133. Ye S, Muntner P, Shimbo D, et al. Behavioral mechanisms, elevated depressive symptoms, and the risk for myocardial infarction or death in individuals with coronary heart disease: the REGARDS (Reason for Geographic and Racial Differences in Stroke) study. *J Am Coll Cardiol.* Feb 12 2013;61(6):622-630.
- 134. Carney RM, Freedland KE, Stein PK, Skala JA, Hoffman P, Jaffe AS. Change in heart rate and heart rate variability during treatment for depression in patients with coronary heart disease. *Psychosom Med.* 2000;62(5):639-647.
- 135. Balogh S, Fitzpatrick DF, Hendricks SE, Paige SR. Increases in heart rate variability with successful treatment in patients with major depressive disorder. *Psychopharmacology Bulletin*. 1993;29(2):201-206.

- 136. Khaykin Y, Dorian P, Baker B, et al. Autonomic correlates of antidepressant treatment using heart-rate variability analysis. *Canadian Journal of Psychiatry Revue Canadienne de Psychiatrie.* 1998;43(2):183-186.
- 137. McFarlane A, Kamath MV, Fallen EL, Malcolm V, Cherian F, Norman G. Effect of sertraline on the recovery rate of cardiac autonomic function in depressed patients after acute myocardial infarction. *American Heart Journal*. 2001;142(4):617-623.
- 138. Doering LV, Cross R, Vredevoe D, Martinez-Maza O, Cowan MJ. Infection, depression, and immunity in women after coronary artery bypass: a pilot study of cognitive behavioral therapy. *Alternative Therapies in Health & Medicine*. 2007;13(3):18-21.
- 139. Lanquillon S, Krieg JC, Bening-Abu-Shach U, Vedder H. Cytokine production and treatment response in major depressive disorder. *Neuropsychopharmacology*. 2000;22(4):370-379.
- 140. Basterzi AD, Aydemir C, Kisa C, et al. IL-6 levels decrease with SSRI treatment in patients with major depression. *Human Psychopharmacology*. 2005;20(7):473-476.
- 141. Lee SK, Lee HS, Lee TB, et al. The effects of antidepressant treatment on serum cytokines and nutritional status in hemodialysis patients. *Journal of Korean medical science*. 2004;19(3):384-389.
- 142. Leo R, Di Lorenzo G, Tesauro M, et al. Association between enhanced soluble CD40 ligand and proinflammatory and prothrombotic states in major depressive disorder: pilot observations on the effects of selective serotonin reuptake inhibitor therapy. *J Clin Psychiatry*. 2006;67(11):1760-1766.
- 143. Pizzi C, Mancini S, Angeloni L, Fontana F, Manzoli L, Costa GM. Effects of selective serotonin reuptake inhibitor therapy on endothelial function and inflammatory markers in patients with coronary heart disease. *Clinical Pharmacology & Therapeutics*. 2009;86(5):527-532.
- 144. Musselman DL, Marzec UM, Manatunga A, et al. Platelet reactivity in depressed patients treated with paroxetine: preliminary findings. *Arch Gen Psychiatry*. 2000;57(9):875-882.
- 145. Pollock BG, Laghrissi-Thode F, Wagner WR. Evaluation of platelet activation in depressed patients with ischemic heart disease after paroxetine or nortriptyline treatment. *Journal of Clinical Psychopharmacology*. 2000;20(2):137-140.
- 146. Serebruany VL, Glassman AH, Malinin AI, et al. Platelet/endothelial biomarkers in depressed patients treated with the selective serotonin reuptake inhibitor sertraline after acute coronary events: the Sertraline AntiDepressant Heart Attack Randomized Trial (SADHART) Platelet Substudy. *Circulation*. 2003;108(8):939-944.
- 147. von Kanel R. Platelet hyperactivity in clinical depression and the beneficial effect of antidepressant drug treatment: how strong is the evidence? *Acta Psychiatr Scand.* Sep 2004;110(3):163-177.
- 148. Hughes JR, Stead LF, Lancaster T. Antidepressants for smoking cessation.[update of Cochrane Database Syst Rev. 2004;(4):CD000031; PMID: 15494986]. *Cochrane Database of Systematic Reviews*. 2007(1):CD000031.
- 149. Trockel M, Burg M, Jaffe A, Barbour K, Taylor CB. Smoking behavior postmyocardial infarction among ENRICHD trial participants: Cognitive behavior therapy intervention for depression and low perceived social support compared with care as usual. *Psychosom Med.* 2008;70(8):875-882.
- 150. Serebruany VL, Suckow RF, Cooper TB, et al. Relationship between release of platelet/endothelial biomarkers and plasma levels of sertraline and N-desmethylsertraline in acute coronary syndrome patients receiving SSRI treatment for depression. *Am J Psychiatry*. Jun 2005;162(6):1165-1170.
- 151. Elderon L, Whooley MA. Depression and cardiovascular disease. *Prog Cardiovasc Dis.* May-Jun 2013;55(6):511-523.
- Duivis HE, de Jonge P, Penninx BW, Na BY, Cohen BE, Whooley MA. Depressive symptoms, health behaviors, and subsequent inflammation in patients with coronary heart disease: prospective findings from the heart and soul study. *Am J Psychiatry*. Sep 2011;168(9):913-920.
- 153. Hayano J, Yamada M, Sakakibara Y, et al. Short- and long-term effects of cigarette smoking on heart rate variability. *Am J Cardiol.* Jan 1 1990;65(1):84-88.
- 154. O'Connor MF, Bower JE, Cho HJ, et al. To assess, to control, to exclude: Effects of biobehavioral factors on circulating inflammatory markers. *Brain Behav Immun*. 2009;23(7):887-897.
- 155. Rennie KL, Hemingway H, Kumari M, Brunner E, Malik M, Marmot M. Effects of moderate and vigorous physical activity on heart rate variability in a British study of civil servants. *Am J Epidemiol.* Jul 15 2003;158(2):135-143.
- 156. LaRosa JC, He J, Vupputuri S. Effect of statins on risk of coronary disease: a meta-analysis of randomized controlled trials. *JAMA*. 1999;282(24):2340-2346.

- 157. Ridker PM. Rosuvastatin in the primary prevention of cardiovascular disease among patients with low levels of low-density lipoprotein cholesterol and elevated high-sensitivity C-reactive protein: rationale and design of the JUPITER trial. *Circulation*. Nov 11 2003;108(19):2292-2297.
- 158. Kroenke K, Spitzer RL, Williams JB. The PHQ-9: Validity of a brief depression severity measure. *Journal of General Internal Medicine*. 2001;16:606-613.
- 159. Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. *J Gen Intern Med.* Nov 2007;22(11):1596-1602.
- 160. Kroenke K, Spitzer RL. The PHQ-9: A new depression diagnostic and severity measure. *Psychiatric Annals*. 2002;32(9):509-515.
- 161. Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. *CMAJ*. Feb 21 2012;184(3):E191-196.
- 162. Wittkampf KA, Naeije L, Schene AH, Huyser J, van Weert HC. Diagnostic accuracy of the mood module of the Patient Health Questionnaire: a systematic review. *Gen Hosp Psychiatry*. Sep-Oct 2007;29(5):388-395.
- 163. Huffman JC, Mastromauro CA, Beach SR, et al. Collaborative Care for Depression and Anxiety Disorders in Patients With Recent Cardiac Events: The Management of Sadness and Anxiety in Cardiology (MOSAIC) Randomized Clinical Trial. *JAMA Intern Med.* Jun 1 2014;174(6):927-936.
- 164. D'Agostino RB, Sr., Vasan RS, Pencina MJ, et al. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. *Circulation*. Feb 12 2008;117(6):743-753.
- 165. Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. *Medical Care*. 2002;40(9):771-781.
- 166. McDonald CJ, Overhage JM, Tierney WM, et al. The Regenstrief Medical Record System: a quarter century experience. *International Journal of Medical Informatics*. 1999;54(3):225-253.
- 167. Davis CD. Prerandomization compliance screening: A statistician's view. In: Shumaker SA, Schron EB, Ockene JK, eds. *The Handbook of Health Behavior Change*. New York: Springer Publishing Company; 1990;342-347.
- 168. Inc. SI. SAS/STAT® 9.2 User's Guide. Cary, NC: SAS Institute Inc.; 2008.
- 169. Hashimoto M, Akishita M, Eto M, et al. Modulation of endothelium-dependent flow-mediated dilatation of the brachial artery by sex and menstrual cycle. *Circulation*. 1995;92(12):3431-3435.
- 170. Moens AL, Goovaerts I, Claeys MJ, Vrints CJ. Flow-mediated vasodilation: a diagnostic instrument, or an experimental tool? *Chest.* 2005;127(6):2254-2263.
- 171. Kaplan GA, Keil JE. Socioeconomic factors and cardiovascular disease: a review of the literature. *Circulation*. Oct 1993;88(4 Pt 1):1973-1998.
- 172. Arean PA, Hegel MT, Unutzer J. *Problem-Solving Therapy for Older Primary Care Patients: Maintenance Group Manual for Project IMPACT.* Los Angeles: University of California Los Angeles; 1999.
- 173. Arean PA, Hegel MT, Unutzer J. *Problem-Solving Treatment in Primary Care: Addendum to PST-PC Treatment Manual for Project IMPACT.* Los Angeles: University of California Los Angeles; 1999.
- 174. Catalan J, Gath DH, Anastasiades P, Bond SA, Day A, Hall L. Evaluation of a brief psychological treatment for emotional disorders in primary care. *Psychological Medicine*. 1991;21(4):1013-1018.
- 175. Hegel MT, Barrett JE, Oxman TE. Training therapists in problem-solving treatment of depressive disorders in primary care: Lessons learned from the treatment effectiveness project. *Families, Systems, & Health.* 2000;18:133-145.
- 176. Hegel MT, Barrett JE, Oxman TE, al. e. *Problem-Solving Treatment for Primary Care (PST-PC): A Treatment Manual for Depression.* Hanover, NH: Dartmouth University; 1999.
- 177. Mynors-Wallis LM, Gath DH, Day A, Baker F. Randomised controlled trial of problem solving treatment, antidepressant medication, and combined treatment for major depression in primary care. *BMJ*. 2000;320(7226):26-30.
- 178. Mago R, Tripathi N, Andrade C. Cardiovascular adverse effects of newer antidepressants. *Expert Rev Neurother*. May 2014;14(5):539-551.
- 179. Mavrides N, Nemeroff CB. Treatment of affective disorders in cardiac disease. *Dialogues Clin Neurosci.* Jun 2015;17(2):127-140.
- 180. Callahan CM. Quality improvement research on late life depression in primary care. *Medical Care*. 2001;39(8):772-784.

- 181. Stein JH, Klein MA, Bellehumeur JL, et al. Use of human immunodeficiency virus-1 protease inhibitors is associated with atherogenic lipoprotein changes and endothelial dysfunction. *Circulation*. Jul 17 2001;104(3):257-262.
- 182. Kathiresan S, Gona P, Larson MG, et al. Cross-sectional relations of multiple biomarkers from distinct biological pathways to brachial artery endothelial function. *Circulation*. Feb 21 2006;113(7):938-945.
- 183. Yeboah J MRLPTS, et al. COmparison of novel risk markers for improvement in cardiovascular risk assessment in intermediate-risk individuals. *JAMA: The Journal of the American Medical Association*. 2012;308(8):788-795.
- 184. Anonymous. Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. *Circulation*. 1996;93:1043-1065.
- 185. Berntson GG, Bigger J, Jr., Eckberg DL, et al. Heart rate variability: Origins, methods, and interpretive caveats. *Psychophysiology*. Nov 1997;34(6):623-648.
- 186. Hawkins MA, Stewart JC, Fitzgerald GJ, Kim S. Combined effect of depressive symptoms and hostility on autonomic nervous system function. *Int J Psychophysiol*. Sep 2011;81(3):317-323.
- 187. Qu MH, Zhang YJ, Webster JG, Tompkins WJ. Motion artifact from spot and band electrodes during impedance cardiography. *IEEE Transactions on Biomedical Engineering*. 1986;33(11):1029-1036.
- 188. Grossman P, Kollai M. Respiratory sinus arrhythmia, cardiac vagal tone, and respiration: within- and between-individual relations. *Psychophysiology*. 1993;30(5):486-495.
- 189. Ernst JM, Litvack DA, Lozano DL, Cacioppo JT, Berntson GG. Impedance pneumography: noise as signal in impedance cardiography. *Psychophysiology*. 1999;36(3):333-338.
- 190. Reed GL. Platelet secretion. In: Michelson AD, ed. *Platelets*. San Diego, CA: Academic Press; 2002.
- 191. Katon W, Von Korff M, Lin E, et al. Stepped collaborative care for primary care patients with persistent symptoms of depression: A randomized trial. *Arch Gen Psychiatry*. 1999;56(12):1109-1115.
- 192. Derogatis LR, Lipman RS, Covi L. SCL-90: an outpatient psychiatric rating scale--preliminary report. *Psychopharmacology Bulletin.* 1973;9(1):13-28.
- 193. Katon W, Robinson P, Von Korff M, et al. A multifaceted intervention to improve treatment of depression in primary care. *Arch Gen Psychiatry*. 1996;53(10):924-932.
- 194. Katon W, Von Korff M, Lin E, et al. Collaborative management to achieve treatment guidelines. Impact on depression in primary care. *JAMA*. 1995;273(13):1026-1031.
- 195. Ridker PM, Danielson E, Fonseca FA, et al. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. *N Engl J Med.* Nov 20 2008;359(21):2195-2207.
- 196. Craig CL, Marshall AL, Sjostrom M, et al. International physical activity questionnaire: 12-country reliability and validity. *Medicine & Science in Sports & Exercise*. 2003;35(8):1381-1395.
- 197. Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. *Medical Care*. 1986;24(1):67-74.
- 198. Nelson DE, Holtzman D, Bolen J, Stanwyck CA, Mack KA. Reliability and validity of measures from the Behavioral Risk Factor Surveillance System (BRFSS). *Social and Preventive Medicine*. 2001;46 Suppl 1:S3-42.
- 199. Perloff D, Grim C, Flack J, et al. Human blood pressure determination by sphygmomanometry. *Circulation*. 1993;88(5):2460-2470.
- 200. Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. *Archives of Internal Medicine*. 2006;166(10):1092-1097.
- 201. Buss AH, Perry M. The aggression questionnaire. *Journal of Personality and Social Psychology*. Sep 1992;63(3):452-459.
- 202. Watson D, Clark LA. *The PANAS-X: Manual for the Positive and Negative Affect Schedule-Expanded Form.* Ames: University of Iowa; 1994.
- 203. Buysse DJ, Reynolds CF, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh sleep quality index: A new instrument for psychiatric practice and research. *Psychiatry research*. 1989;28:193-213.
- 204. Mason MJ. A review of procedural and statistical methods for handling attrition and missing data. *Measurement and Evaluation in Counseling and Development*. 1999;32:111-118.
- 205. Blumenthal JA, Sherwood A, Babyak MA, et al. Effects of exercise and stress management training on markers of cardiovascular risk in patients with ischemic heart disease: a randomized controlled trial. *JAMA*. 2005;293(13):1626-1634.

- 206. Paul-Labrador M, Polk D, Dwyer JH, et al. Effects of a randomized controlled trial of transcendental meditation on components of the metabolic syndrome in subjects with coronary heart disease. *Archives of Internal Medicine*. 2006;166(11):1218-1224.
- 207. van Dixhoorn J. Cardiorespiratory effects of breathing and relaxation instruction in myocardial infarction patients. *Biol Psychol.* 1998;49(1-2):123-135.
- 208. Fisher L, Dixon D, Herson J, Frankowski R, Hearon M, Pearce K. Intention to treat in clinical trials. In: Pearce K, ed. *Statistical Issues in Drug Research and Development*. New York: Marcel Kekker; 1990:331-350.
- 209. MacKinnon DP, Fairchild AJ. Current directions in mediation analysis. *Current Directions in Psychological Science*. 2009;18(1):16-20.
- 210. MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. *Psychological Methods*. 2002;7:83-104.